CLINICAL TRIAL: NCT03275389
Title: Reactogenicity, Safety and Immunogenicity Study of GlaxoSmithKline (GSK) Biologicals' Investigational Supra-seasonal Universal Influenza Vaccines - Inactivated (SUIVs) (GSK3816302A) in Healthy Adults
Brief Title: A Study to Evaluate the Reactogenicity, Safety and Immunogenicity of GlaxoSmithKline (GSK) Biologicals' Investigational Supra-seasonal Universal Influenza Vaccines - Inactivated (SUIVs) (GSK3816302A) in Healthy Adults Aged 18 to 39 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 207543; 2017-001584-20 (EudraCT Number)
Record Dates: First submitted 2017-08-29; First posted 2017-09-07 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Influenza, Human
Keywords: Safety; Healthy adults; Immunogenicity; Supra-seasonal universal influenza vaccines - inactivated (SUIVs)
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The site staff will work in an observer-blind manner. As the vaccines appearance and preparation are different, two teams of study personnel will be set up:
  * A team of unblinded personnel (responsible for the reception, preparation and administration of the vaccines).
  * A team of blinded personnel (responsible for the clinical safety evaluation of the subjects).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- D-SUIV Adjuvanted Group 1 (Experimental): Subjects received one dose of D-SUIV cH8/1N1+AS03 vaccine at Day 1, one dose of Placebo at Day 57 and one booster dose of D-SUIV cH5/1N1+AS03 vaccine at Month 14. All doses were administered intramuscularly in the non-dominant arm.
  Interventions: Biological: D-SUIV cH8/1N1+AS03; Biological: D-SUIV cH5/1N1+AS03; Biological: Placebo
- D-SUIV Adjuvanted Group 2 (Experimental): Subjects received one dose of D-SUIV cH5/1N1+AS03 vaccine at Day 1, one dose of Placebo at Day 57 and one booster dose of D-SUIV cH8/1N1+AS03 vaccine at Month 14. All doses were administered intramuscularly in the non-dominant arm.
  Interventions: Biological: D-SUIV cH8/1N1+AS03; Biological: D-SUIV cH5/1N1+AS03; Biological: Placebo
- D-SUIV Adjuvanted Group 3 (Experimental): Subjects received one dose of D-SUIV cH8/1N1+AS03 vaccine at Day 1, one dose D-SUIV cH5/1N1+AS03 vaccine at Day 57 and one booster dose of D-SUIV cH11/1N1+AS03 vaccine at Month 14. All doses were administered intramuscularly in the non-dominant arm.
  Interventions: Biological: D-SUIV cH8/1N1+AS03; Biological: D-SUIV cH5/1N1+AS03; Biological: D-SUIV cH11/1N1+AS03
- D-SUIV Adjuvanted Group 4 (Experimental): Subjects received one dose of D-SUIV cH8/1N1+AS01 vaccine at Day 1, one dose of Placebo at Day 57 and one booster dose of D-SUIV cH5/1N1+AS01 vaccine at Month 14. All doses were administered intramuscularly in the non-dominant arm.
  Interventions: Biological: D-SUIV cH8/1N1+AS01; Biological: D-SUIV cH5/1N1+AS01; Biological: Placebo
- D-SUIV Adjuvanted Group 5 (Experimental): Subjects received one dose of D-SUIV cH5/1N1+AS01 vaccine at Day 1, one dose of Placebo at Day 57 and one booster dose of D-SUIV cH8/1N1+AS01 vaccine at Month 14. All doses were administered intramuscularly in the non-dominant arm.
  Interventions: Biological: D-SUIV cH8/1N1+AS01; Biological: D-SUIV cH5/1N1+AS01; Biological: Placebo
- D-SUIV Adjuvanted Group 6 (Experimental): Subjects received one dose of D-SUIV cH8/1N1+AS01 vaccine at Day 1, one dose of D-SUIV cH5/1N1+AS01 vaccine at Day 57 and one booster dose of D-SUIV cH11/1N1+AS01 vaccine at Month 14. All doses were administered intramuscularly in the non-dominant arm.
  Interventions: Biological: D-SUIV cH8/1N1+AS01; Biological: D-SUIV cH5/1N1+AS01; Biological: D-SUIV cH11/1N1+AS01
- D-SUIV Unadjuvanted Group 1 (Experimental): Subjects received one dose of D-SUIV cH8/1N1 vaccine at Day 1, one dose of Placebo at Day 57 and one booster dose of D-SUIV cH5/1N1 vaccine at Month 14. All doses were administered intramuscularly in the non-dominant arm.
  Interventions: Biological: D-SUIV cH8/1N1; Biological: D-SUIV cH5/1N1; Biological: Placebo
- D-SUIV Unadjuvanted Group 2 (Experimental): Subjects received one dose of D-SUIV cH5/1N1 vaccine at Day 1, one dose of Placebo at Day 57 and one booster dose of D-SUIV cH8/1N1 vaccine at Month 14. All doses were administered intramuscularly in the non-dominant arm.
  Interventions: Biological: D-SUIV cH8/1N1; Biological: D-SUIV cH5/1N1; Biological: Placebo
- D-SUIV Unadjuvanted Group 3 (Experimental): Subjects received one dose of D-SUIV cH8/1N1 vaccine at Day 1, one dose of D-SUIV cH5/1N1 vaccine at Day 57 and one booster dose of D-SUIV cH11/1N1 vaccine at Month 14. All doses were administered intramuscularly in the non-dominant arm.
  Interventions: Biological: D-SUIV cH8/1N1; Biological: D-SUIV cH5/1N1; Biological: D-SUIV cH11/1N1
- IIV4 Group (Active Comparator): Subjects received one dose of Fluarix Quadrivalent (IIV4) vaccine at Day 1, one dose of Placebo at Day 57 and one dose of Fluarix Quadrivalent vaccine at Month 14. All doses were administered intramuscularly in the non-dominant arm.
  Interventions: Biological: Placebo; Biological: Fluarix Quadrivalent

INTERVENTIONS:
Biological: D-SUIV cH8/1N1+AS03 — 1 Primary dose or 1 Booster dose of Supraseasonal Universal Influenza Vaccine (Flu D-SUIV), chimeric strain cH8/1N1 with Adjuvant System 03 (AS03) was administered intramuscularly (IM) in the deltoid region of non-dominant arm.
  Arms: D-SUIV Adjuvanted Group 1; D-SUIV Adjuvanted Group 2; D-SUIV Adjuvanted Group 3
Biological: D-SUIV cH5/1N1+AS03 — 1 Primary dose or 1 Booster dose of Supraseasonal Universal Influenza Vaccine (Flu D-SUIV), chimeric strain cH5/1N1 with Adjuvant System 03 (AS03) was administered IM in the deltoid region of non-dominant arm.
  Arms: D-SUIV Adjuvanted Group 1; D-SUIV Adjuvanted Group 2; D-SUIV Adjuvanted Group 3
Biological: D-SUIV cH11/1N1+AS03 — 1 Booster dose of Supraseasonal Universal Influenza Vaccine (Flu D-SUIV), chimeric strain cH11/1N1 with Adjuvant System 03 (AS03) was administered IM in the deltoid region of non-dominant arm.
  Arms: D-SUIV Adjuvanted Group 3
Biological: D-SUIV cH8/1N1+AS01 — 1 Primary dose or 1 Booster dose of Supraseasonal Universal Influenza Vaccine (Flu D-SUIV), chimeric strain cH8/1N1 with Adjuvant System 01 (AS01) was administered IM in the deltoid region of non-dominant arm.
  Arms: D-SUIV Adjuvanted Group 4; D-SUIV Adjuvanted Group 5; D-SUIV Adjuvanted Group 6
Biological: D-SUIV cH5/1N1+AS01 — 1 Primary dose or 1 Booster dose of Supraseasonal Universal Influenza Vaccine (Flu D-SUIV), chimeric strain cH5/1N1 with Adjuvant System 01 (AS01) was administered IM in the deltoid region of non-dominant arm.
  Arms: D-SUIV Adjuvanted Group 4; D-SUIV Adjuvanted Group 5; D-SUIV Adjuvanted Group 6
Biological: D-SUIV cH11/1N1+AS01 — 1 Booster dose of Supraseasonal Universal Influenza Vaccine (Flu D-SUIV), chimeric strain cH11/1N1 with Adjuvant System 01 (AS01) was administered IM in the deltoid region of non-dominant arm.
  Arms: D-SUIV Adjuvanted Group 6
Biological: D-SUIV cH8/1N1 — 1 Primary dose or 1 Booster dose of Supraseasonal Universal Influenza Vaccine (Flu D-SUIV), chimeric strain cH8/1N1 without adjuvant was administered IM in the deltoid region of non-dominant arm.
  Arms: D-SUIV Unadjuvanted Group 1; D-SUIV Unadjuvanted Group 2; D-SUIV Unadjuvanted Group 3
Biological: D-SUIV cH5/1N1 — 1 Primary dose or 1 Booster dose of Supraseasonal Universal Influenza Vaccine (Flu D-SUIV), chimeric strain cH5/1N1 without adjuvant was administered IM in the deltoid region of non-dominant arm.
  Arms: D-SUIV Unadjuvanted Group 1; D-SUIV Unadjuvanted Group 2; D-SUIV Unadjuvanted Group 3
Biological: D-SUIV cH11/1N1 — 1 Booster dose of Supraseasonal Universal Influenza Vaccine (Flu D-SUIV), chimeric strain cH11/1N1 without adjuvant was administered IM in the deltoid region of non-dominant arm.
  Arms: D-SUIV Unadjuvanted Group 3
Biological: Placebo — 1 dose of Phosphate Buffered Saline (PBS) was administered IM in the deltoid region of non-dominant arm.
  Arms: D-SUIV Adjuvanted Group 1; D-SUIV Adjuvanted Group 2; D-SUIV Adjuvanted Group 4; D-SUIV Adjuvanted Group 5; D-SUIV Unadjuvanted Group 1; D-SUIV Unadjuvanted Group 2; IIV4 Group
Biological: Fluarix Quadrivalent — 1 Primary dose and 1 Booster dose was administered IM in the deltoid region of non-dominant arm.
  Arms: IIV4 Group

SUMMARY:
The purpose of this study is to assess the reactogenicity, safety and immunogenicity of different formulations of GlaxoSmithKline (GSK) Biologicals' investigational supra-seasonal universal influenza vaccines (SUIVs) (unadjuvanted or adjuvanted) in 18 to 39 year-old healthy subjects. Subjects will be enrolled and vaccinated with one or 2 primary dose(s) followed by a booster dose one year later.

DETAILED DESCRIPTION:
Current seasonal influenza vaccines show good efficacy when they are well-matched with the circulating virus strains.

However, influenza viruses constantly change their surface glycoproteins that are the targets of most immune responses, allowing them to escape pre-existing immunity, a process called antigenic drift. Therefore, seasonal influenza vaccines have to be reformulated and re-administered on an annual basis. In addition, novel viruses can appear at irregular intervals and cause influenza virus pandemics that can claim millions of lives.

GSK Biologicals is now developing a new influenza vaccine that contains modified inactivated influenza viruses. The purpose of this approach is to elicit an immune response that would protect against all current and future circulating influenza strains without having to administer the vaccine each year.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performance of any study specific procedure.
* A male or female between, and including, 18 and 39 years of age at the time of the first vaccination.
* Healthy subjects without acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as established by medical history and clinical examination before first vaccination and laboratory screening tests (the latter being only applicable for subjects enrolled in Phase I).
* Subjects with no history of influenza vaccination within 6 months prior to first study vaccination and who are willing to forego any influenza vaccination during the entire study period.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * Has practiced adequate contraception for 30 days prior to first vaccination, and
  * Has a negative pregnancy test on the day of vaccination, and
  * Has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series (last vaccination at Month 14).

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines during the period starting 30 days before the first dose of study vaccines, or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting 6 months prior to the first vaccine dose. For corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs within 6 months before first vaccination, or planned administration any time during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose up to the blood sampling at Day 85 and in the period starting 30 days before booster vaccination at Month 14 up to the blood sample at Month 14 + 28 days.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Previous vaccination against influenza within the 6 months preceding the first vaccination at Visit 1 or planned use of such vaccines during the study period.
* History of vaccination with a (pre)pandemic influenza vaccine other than an H1N1pdm09 vaccine or history of laboratory-confirmed influenza infection other than seasonal or H1N1pdm09 influenza.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of or current autoimmune disease.
* Subjects diagnosed with excessive daytime sleepiness or narcolepsy; or history of narcolepsy in a subject's parent or sibling.
* History of Guillain-Barré syndrome.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Hypersensitivity to latex.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 38.0°C / 100.4°F. The preferred location for measuring temperature in this study will be the oral cavity.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
  * For subjects with acute disease and/or fever at the time of enrolment, Visit 1 may be re-scheduled within the allowed time-window.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the first dose of study vaccines or planned administration during the study period.
* Blood donation within 30 days before the first study blood sampling or planned blood donation within 30 days before and up to 30 days after any study blood sampling.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Additional criterion applicable for Phase I subjects:

* Hematological and/or biochemical parameters outside the laboratory normal ranges, unless the laboratory abnormalities are considered not clinically significant by the investigator.
* Liver enzymes (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]) outside of the normal laboratory ranges.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 470 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (5):
  - GSK Investigational Site, South Miami, Florida
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Norfolk, Virginia
- GSK Investigational Site, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Folschweiller N, Vanden Abeele C, Chu L, Van Damme P, Garcia-Sastre A, Krammer F, Nachbagauer R, Palese P, Solorzano A, Bi D, David MP, Friel D, Innis BL, Koch J, Mallett CP, Rouxel RN, Salaun B, Vantomme V, Verheust C, Struyf F. Reactogenicity, safety, and immunogenicity of chimeric haemagglutinin influenza split-virion vaccines, adjuvanted with AS01 or AS03 or non-adjuvanted: a phase 1-2 randomised controlled trial. Lancet Infect Dis. 2022 Jul;22(7):1062-1075. doi: 10.1016/S1473-3099(22)00024-X. Epub 2022 Apr 21. PMID 35461522

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 470 subjects were enrolled and randomized in the study, however, while 2 subjects were allocated subjects numbers, they did not receive any vaccine dose.
Period: Overall Study
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Started | 45 | 46 | 47 | 47 | 48 | 47 | 47 | 48 | 46 | 47
Completed | 34 | 30 | 24 | 25 | 32 | 29 | 22 | 30 | 31 | 29
Not Completed | 11 | 16 | 23 | 22 | 16 | 18 | 25 | 18 | 15 | 18
Not completed — Lost to Follow-up | 10 | 10 | 19 | 12 | 11 | 12 | 21 | 15 | 12 | 14
Not completed — SERIOUS ADVERSE EVENT AND/OR PIMD | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — CONSENT WITHDRAWAL NOT DUE TO ADV. EVENT | 1 | 0 | 0 | 5 | 3 | 3 | 3 | 3 | 2 | 2
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — NOT WILLING TO PARTICIPATE THIS VISIT | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 4 | 3 | 2 | 2 | 2 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group | Total
Number analyzed (Participants) | 45 | 46 | 47 | 47 | 48 | 47 | 47 | 48 | 46 | 47 | 468
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.0 (6.6) | 29.3 (5.7) | 28.6 (6.0) | 28.7 (6.4) | 29.1 (6.2) | 28.8 (6.1) | 29.6 (5.8) | 28.5 (5.9) | 28.8 (5.9) | 29.3 (5.8) | 29.0 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 28 | 28 | 27 | 27 | 27 | 26 | 25 | 27 | 268
  Male | 19 | 19 | 19 | 19 | 21 | 20 | 20 | 22 | 21 | 20 | 200
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American indian or alaska native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian - central / south asian heritage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian - east asian heritage | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian - south east asian heritage | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Black or african american | 11 | 9 | 10 | 8 | 5 | 7 | 10 | 13 | 6 | 9 | 88
  Native hawaiian or other pacific islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Other, Not specified | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 2 | 1 | 10
  White - arabic / north african heritage | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 5
  White - caucasian / european heritage | 34 | 34 | 37 | 36 | 40 | 38 | 35 | 33 | 37 | 35 | 359

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Solicited Local Adverse Events (AEs) After First Dose Administration
Description: Assessed solicited local symptoms are pain, erythema and swelling. Any = occurrence of the symptom regardless of intensity grade. Any erythema/swelling = erythema/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 1-7) follow-up period after first vaccine dose
Population: Analysis was performed on the Exposed Set (ES) which included all subjects with the vaccine dose documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 46 | 45 | 47 | 46 | 45
Participants
  Erythema | 1 | 3 | 2 | 2 | 1 | 3 | 1 | 0 | 1 | 0
  Pain | 34 | 42 | 37 | 39 | 40 | 42 | 16 | 13 | 15 | 35
  Swelling | 4 | 2 | 2 | 4 | 3 | 2 | 0 | 0 | 1 | 0

2. Primary Outcome: Number of Subjects With Solicited Local AEs After Second Dose Administration
Description: as for outcome 1
Time Frame: During the 7-day (Days 1-7) follow-up period after second vaccine dose
Population: Analysis was performed on the ES which included all subjects with the vaccine dose documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 40 | 37 | 36 | 41 | 41 | 37 | 38 | 39 | 40 | 39
Participants
  Erythema | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain | 5 | 2 | 29 | 2 | 8 | 32 | 4 | 5 | 12 | 10
  Swelling | 0 | 0 | 4 | 0 | 0 | 2 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Subjects With Solicited Local AEs After Booster Dose Administration
Description: Assessed solicited local symptoms are pain, erythema and swelling. Any = occurrence of the symptom regardless of intensity grade. Any erythema/swelling = erythema/swelling spreading beyond 20 mm of injection site.
Time Frame: During the 7-day (Days 1-7) follow-up period after booster vaccine dose
Population: Analysis was performed on the ES which included all subjects with the vaccine dose documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 33 | 32 | 27 | 30 | 31 | 30 | 24 | 32 | 33 | 31
Participants
  Erythema | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Pain | 27 | 31 | 26 | 29 | 28 | 25 | 4 | 10 | 13 | 21
  Swelling | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Subjects With Solicited General AEs After First Dose Administration
Description: Assessed solicited general symptoms are arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, shivering and fever [defined as oral temperature equal to or above 38.0 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade
Time Frame: During the 7-day (Days 1-7) follow-up period after first vaccine dose
Population: Analysis was performed on the ES which included all subjects with the vaccine dose documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 46 | 45 | 47 | 46 | 46
Participants
  Arthralgia | 4 | 6 | 9 | 2 | 3 | 8 | 6 | 5 | 2 | 5
  Fatigue | 17 | 18 | 22 | 18 | 21 | 18 | 17 | 19 | 12 | 12
  Gastrointestinal symptoms | 6 | 7 | 10 | 6 | 8 | 8 | 6 | 8 | 10 | 8
  Headache | 18 | 18 | 19 | 23 | 16 | 26 | 16 | 19 | 15 | 14
  Myalgia | 16 | 13 | 19 | 17 | 19 | 20 | 9 | 9 | 6 | 11
  Shivering | 6 | 3 | 10 | 10 | 8 | 9 | 2 | 2 | 2 | 3
  Temperature | 1 | 1 | 0 | 2 | 2 | 1 | 1 | 1 | 0 | 0

5. Primary Outcome: Number of Subjects With Solicited General AEs After Second Dose Administration
Description: as for outcome 4
Time Frame: During the 7-day (Days 1-7) follow-up period after second vaccine dose
Population: Analysis was performed on the ES which included all subjects with the vaccine dose documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 40 | 37 | 36 | 41 | 41 | 39 | 38 | 39 | 40 | 40
Participants
  Arthralgia | 3 | 4 | 4 | 0 | 4 | 4 | 0 | 0 | 2 | 2
  Fatigue | 7 | 7 | 10 | 6 | 7 | 8 | 5 | 5 | 10 | 5
  Gastrointestinal symptoms | 3 | 4 | 4 | 3 | 3 | 6 | 1 | 4 | 2 | 2
  Headache | 8 | 12 | 13 | 7 | 9 | 12 | 5 | 12 | 8 | 7
  Myalgia | 5 | 6 | 12 | 1 | 4 | 16 | 3 | 2 | 6 | 3
  Shivering | 2 | 4 | 4 | 0 | 3 | 5 | 1 | 0 | 2 | 1
  Temperature | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Subjects With Solicited General AEs After Booster Dose Administration
Description: as for outcome 4
Time Frame: During the 7-day (Days 1-7) follow-up period after booster vaccine dose
Population: Analysis was performed on the ES which included all subjects with the vaccine dose documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 33 | 32 | 27 | 30 | 31 | 30 | 24 | 32 | 33 | 31
Participants
  Arthralgia | 6 | 8 | 4 | 4 | 9 | 4 | 1 | 1 | 2 | 1
  Fatigue | 15 | 19 | 17 | 16 | 20 | 9 | 2 | 6 | 6 | 3
  Gastrointestinal symptoms | 3 | 8 | 8 | 5 | 6 | 5 | 1 | 2 | 4 | 0
  Headache | 9 | 13 | 14 | 15 | 16 | 15 | 3 | 7 | 6 | 4
  Myalgia | 15 | 17 | 15 | 15 | 13 | 10 | 0 | 4 | 5 | 3
  Shivering | 5 | 13 | 6 | 6 | 14 | 9 | 0 | 1 | 2 | 1
  Temperature | 2 | 3 | 1 | 4 | 2 | 1 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Subjects With Any Unsolicited AEs Post-vaccination Period
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any is defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination
Time Frame: During the 28-day (Days 1-28) follow-up period accross doses
Population: Analysis was performed on the ES which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 45 | 46 | 47 | 47 | 48 | 47 | 47 | 48 | 46 | 47
Participants | 27 | 23 | 23 | 24 | 24 | 17 | 22 | 23 | 22 | 21

8. Primary Outcome: Number of Subjects With Change From Baseline in Hematological and Biochemical Laboratory Results at Day 8 by Toxicity Grading
Description: Hematological parameters assessed are: Eosinophils increase [EOSi], hemoglobin decrease [HEMd] , lymphocytes decrease [LYMd], Neutrophils decrease [NEUd], platelets decrease [PLTCd], white blood cells decrease [WBCd], WBC increase [WBCi]. Biochemical parameters assessed are: alanine aminotransferase increase [ALTi], aspartate aminotransferase increase [ASTi], blood urea nitrogen [BUN], creatinine [CRE].Toxicity grading is according to the Food and Drug Administration (FDA) guidance for industry: Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical Trials (September 2007). The grading scale is defined as follows: mild (Grade 1), moderate (Grade 2), severe (Grade 3) and potentially life threatening (Grade 4). Category naming has been defined as follows: Parameter- grading at Baseline- grading at Timing: e.g.: "ALT-Grade 0-Grade 1".
Time Frame: At Day 8
Population: Analysis was performed on the ES which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 45 | 46
Participants
  ALTi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALTi, GRADE 0, UNKNOWN: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1
  ALTi, GRADE 0, GRADE 0: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 0 | 40 | 45 | 42 | 41 | 45 | 45 | 43 | 44 | 41 | 44
  ALTi, GRADE 0, GRADE 1: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  ALTi, GRADE 0, GRADE 3: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ALTi, GRADE 1, GRADE 0: number analyzed (Participants) | 4 | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 0
  ALTi, GRADE 1, GRADE 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 0
  ALTi, GRADE 1, GRADE 1: number analyzed (Participants) | 4 | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 0
  ALTi, GRADE 1, GRADE 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  ASTi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ASTi, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ASTi, GRADE 0, UNKNOWN: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1
  ASTi, GRADE 0, GRADE 0: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 0 | 44 | 46 | 44 | 42 | 46 | 45 | 42 | 44 | 44 | 44
  ASTi, GRADE 0, GRADE 1: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  ASTi, GRADE 0, GRADE 2: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  ASTi, GRADE 0, GRADE 4: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ASTi, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  ASTi, GRADE 1, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  ASTi, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ASTi, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  BUN, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  BUN, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  BUN, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, UNKNOWN | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1
  BUN, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 0 | 43 | 46 | 45 | 43 | 46 | 46 | 43 | 47 | 43 | 45
  BUN, GRADE 1, GRADE 0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 1, GRADE 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  CRE, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  CRE, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  CRE, GRADE 0, UNKNOWN | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1
  CRE, GRADE 0, GRADE 0 | 44 | 46 | 45 | 43 | 46 | 46 | 43 | 47 | 45 | 45
  EOSi, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  EOSi, UNKNOWN, GRADE 0 | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  EOSi, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, UNKNOWN | 2 | 0 | 2 | 1 | 0 | 0 | 2 | 2 | 1 | 2
  EOSi, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, GRADE 0 | 41 | 43 | 38 | 43 | 45 | 44 | 40 | 43 | 38 | 41
  EOSi, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, GRADE 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0
  EOSi, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  EOSi, GRADE 1, GRADE 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  EOSi, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  EOSi, GRADE 1, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  HEMd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  HEMd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  HEMd, GRADE 0, UNKNOWN: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, UNKNOWN | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 2
  HEMd, GRADE 0, GRADE 0: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 0 | 37 | 37 | 40 | 39 | 43 | 40 | 37 | 40 | 40 | 40
  HEMd, GRADE 0, GRADE 1: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 1 | 1 | 4 | 1 | 1 | 1 | 3 | 1 | 1 | 2 | 1
  HEMd, GRADE 0, GRADE 2: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  HEMd, GRADE 1, UNKNOWN: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  HEMd, GRADE 1, GRADE 0: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
  HEMd, GRADE 1, GRADE 1: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 1 | 3 | 1 | 2 | 4 | 0 | 1 | 2 | 0 | 0 | 0
  HEMd, GRADE 1, GRADE 2: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  HEMd, GRADE 2, GRADE 1: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0
  HEMd, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  HEMd, GRADE 2, GRADE 2: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0
  HEMd, GRADE 2, GRADE 2 | 2 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 0
  HEMd, GRADE 2, GRADE 3: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0
  HEMd, GRADE 2, GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  HEMd, GRADE 3, UNKNOWN: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  HEMd, GRADE 3, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  HEMd, GRADE 3, GRADE 3: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  HEMd, GRADE 3, GRADE 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  LYMd, UNKNOWN, GRADE 0 | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  LYMd, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, UNKNOWN | 2 | 0 | 2 | 1 | 0 | 0 | 2 | 2 | 1 | 2
  LYMd, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 0 | 39 | 45 | 37 | 44 | 43 | 45 | 42 | 42 | 38 | 41
  LYMd, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  LYMd, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 2: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NEUd, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 0 | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 2 | 1
  NEUd, UNKNOWN, GRADE 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  NEUd, UNKNOWN, GRADE 2: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  NEUd, GRADE 0, UNKNOWN: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, UNKNOWN | 2 | 0 | 2 | 1 | 0 | 0 | 2 | 2 | 1 | 2
  NEUd, GRADE 0, GRADE 0: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 0 | 37 | 40 | 39 | 41 | 41 | 43 | 39 | 38 | 37 | 37
  NEUd, GRADE 0, GRADE 1: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2
  NEUd, GRADE 0, GRADE 2: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
  NEUd, GRADE 1, GRADE 0: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 0 | 1 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  NEUd, GRADE 1, GRADE 1: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0
  NEUd, GRADE 1, GRADE 2: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  NEUd, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 2, GRADE 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 3, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NEUd, GRADE 3, GRADE 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  PLTCd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  PLTCd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  PLTCd, GRADE 0, UNKNOWN: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, UNKNOWN | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 2 | 1 | 2
  PLTCd, GRADE 0, GRADE 0: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 0 | 43 | 45 | 42 | 43 | 46 | 45 | 42 | 44 | 43 | 43
  PLTCd, GRADE 0, GRADE 1: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  PLTCd, GRADE 0, GRADE 2: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLTCd, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  PLTCd, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  PLTCd, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCd, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, UNKNOWN | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 2 | 1 | 2
  WBCd, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, GRADE 0 | 41 | 45 | 42 | 44 | 44 | 46 | 41 | 42 | 41 | 43
  WBCd, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, GRADE 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  WBCd, GRADE 1, GRADE 0: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0
  WBCd, GRADE 1, GRADE 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0
  WBCd, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBCd, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBCi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCi, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCi, GRADE 0, UNKNOWN: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, UNKNOWN | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 2 | 1 | 2
  WBCi, GRADE 0, GRADE 0: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 0 | 41 | 43 | 42 | 42 | 45 | 45 | 39 | 39 | 38 | 39
  WBCi, GRADE 0, GRADE 1: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 3
  WBCi, GRADE 1, GRADE 0: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0
  WBCi, GRADE 1, GRADE 1: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 1
  WBCi, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCi, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

9. Primary Outcome: Number of Subjects With Change in Hematological and Biochemical Laboratory Results From Day 8 to Day 29 Versus Baseline by Toxicity Grading
Description: Hematological parameters assessed are: EOSi, HEMd, LYMd, NEUd, PLTCd, WBCd, WBCi. Biochemical parameters assessed are: ALTi, ASTi, BUN, CRE. Toxicity grading is according to the FDA guidance for industry: Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical Trials (September 2007). The grading scale is defined as following: mild (Grade 1), moderate (Grade 2), severe (Grade 3) and potentially life threatening (Grade 4). Category naming has been defined as: Parameter-grading at Baseline-grading at Timing: e.g.: "ALT-Grade 0-Grade 1". The reported results consider any change that occurred during the defined time frame: i.e. any abnormality occurring at an intermediate visit leading to a maximum change from baseline, during the period covered, is the reported result for the outcome.
Time Frame: From Day 8 to Day 29
Population: Analysis was performed on the ES which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 45 | 46
Participants
  ALTi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALTi, GRADE 0, UNKNOWN: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALTi, GRADE 0, GRADE 0: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 0 | 40 | 45 | 41 | 44 | 45 | 44 | 41 | 43 | 40 | 44
  ALTi, GRADE 0, GRADE 1: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 1 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 3 | 2
  ALTi, GRADE 0, GRADE 2: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ALTi, GRADE 0, GRADE 3: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ALTi, GRADE 1, GRADE 0: number analyzed (Participants) | 4 | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 0
  ALTi, GRADE 1, GRADE 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 0
  ALTi, GRADE 1, GRADE 1: number analyzed (Participants) | 4 | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 0
  ALTi, GRADE 1, GRADE 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  ASTi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ASTi, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ASTi, GRADE 0, UNKNOWN: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ASTi, GRADE 0, GRADE 0: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 0 | 44 | 46 | 44 | 45 | 46 | 44 | 42 | 43 | 42 | 45
  ASTi, GRADE 0, GRADE 1: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 2 | 0
  ASTi, GRADE 0, GRADE 2: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  ASTi, GRADE 0, GRADE 4: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ASTi, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  ASTi, GRADE 1, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ASTi, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  ASTi, GRADE 1, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  ASTi, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ASTi, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  BUN, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  BUN, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  BUN, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  BUN, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 0 | 43 | 45 | 45 | 46 | 46 | 46 | 43 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, GRADE 1, GRADE 0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 1, GRADE 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  CRE, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  CRE, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  CRE, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  CRE, GRADE 0, GRADE 0 | 44 | 46 | 45 | 46 | 46 | 46 | 43 | 47 | 45 | 46
  EOSi, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  EOSi, UNKNOWN, GRADE 0 | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 2 | 5 | 2
  EOSi, UNKNOWN, GRADE 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  EOSi, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  EOSi, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  EOSi, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, GRADE 0 | 43 | 43 | 40 | 44 | 45 | 44 | 40 | 45 | 39 | 43
  EOSi, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, GRADE 1 | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 0 | 1 | 0
  EOSi, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  EOSi, GRADE 1, GRADE 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  EOSi, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  EOSi, GRADE 1, GRADE 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  HEMd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  HEMd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  HEMd, GRADE 0, GRADE 0: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 0 | 37 | 37 | 41 | 38 | 43 | 40 | 37 | 39 | 39 | 42
  HEMd, GRADE 0, GRADE 1: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 1 | 2 | 4 | 1 | 3 | 1 | 3 | 2 | 3 | 4 | 1
  HEMd, GRADE 0, GRADE 2: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  HEMd, GRADE 1, UNKNOWN: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  HEMd, GRADE 1, GRADE 0: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
  HEMd, GRADE 1, GRADE 1: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 1 | 3 | 1 | 2 | 4 | 0 | 1 | 2 | 0 | 0 | 0
  HEMd, GRADE 1, GRADE 2: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  HEMd, GRADE 2, GRADE 2: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0
  HEMd, GRADE 2, GRADE 2 | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 0
  HEMd, GRADE 2, GRADE 3: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0
  HEMd, GRADE 2, GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  HEMd, GRADE 3, GRADE 3: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  HEMd, GRADE 3, GRADE 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  LYMd, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  LYMd, UNKNOWN, GRADE 0 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  LYMd, UNKNOWN, GRADE 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  LYMd, UNKNOWN, GRADE 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  LYMd, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 0 | 41 | 45 | 39 | 45 | 42 | 45 | 43 | 43 | 39 | 41
  LYMd, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3
  LYMd, GRADE 0, GRADE 2: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 2: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NEUd, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 0 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 2 | 1
  NEUd, UNKNOWN, GRADE 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  NEUd, UNKNOWN, GRADE 2: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  NEUd, GRADE 0, UNKNOWN: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  NEUd, GRADE 0, GRADE 0: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 0 | 38 | 39 | 40 | 40 | 40 | 42 | 37 | 38 | 38 | 38
  NEUd, GRADE 0, GRADE 1: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 1 | 3 | 2 | 1 | 2 | 1 | 1 | 2 | 3 | 0 | 2
  NEUd, GRADE 0, GRADE 2: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 2 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 1 | 1
  NEUd, GRADE 0, GRADE 3: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  NEUd, GRADE 1, GRADE 0: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  NEUd, GRADE 1, GRADE 1: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1
  NEUd, GRADE 1, GRADE 2: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
  NEUd, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 2, GRADE 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  NEUd, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  NEUd, GRADE 2, GRADE 2: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 2, GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  NEUd, GRADE 3, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NEUd, GRADE 3, GRADE 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  PLTCd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  PLTCd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  PLTCd, GRADE 0, UNKNOWN: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  PLTCd, GRADE 0, GRADE 0: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 0 | 43 | 45 | 44 | 44 | 46 | 45 | 43 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 1: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  PLTCd, GRADE 0, GRADE 2: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLTCd, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 2: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  PLTCd, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  PLTCd, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  WBCd, UNKNOWN, GRADE 1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCd, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  WBCd, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WBCd, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, GRADE 0 | 41 | 44 | 44 | 43 | 43 | 46 | 42 | 44 | 41 | 42
  WBCd, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, GRADE 1 | 2 | 1 | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 3
  WBCd, GRADE 1, GRADE 0: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0
  WBCd, GRADE 1, GRADE 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0
  WBCd, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBCd, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBCi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCi, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCi, GRADE 0, UNKNOWN: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WBCi, GRADE 0, GRADE 0: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 0 | 42 | 40 | 43 | 42 | 45 | 45 | 38 | 39 | 39 | 41
  WBCi, GRADE 0, GRADE 1: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 1 | 0 | 3 | 1 | 2 | 0 | 1 | 3 | 5 | 1 | 3
  WBCi, GRADE 1, GRADE 0: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0
  WBCi, GRADE 1, GRADE 1: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 1
  WBCi, GRADE 1, GRADE 2: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBCi, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCi, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

10. Primary Outcome: Number of Subjects With Change in Hematological and Biochemical Laboratory Results From Day 8 to Day 85 Versus Baseline by Toxicity Grading
Description: as for outcome 9
Time Frame: From Day 8 to Day 85
Population: Analysis was performed on the ES which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 45 | 46
Participants
  ALTi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALTi, GRADE 0, UNKNOWN: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALTi, GRADE 0, GRADE 0: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 0 | 39 | 42 | 39 | 42 | 44 | 42 | 39 | 39 | 35 | 43
  ALTi, GRADE 0, GRADE 1: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 1 | 0 | 4 | 4 | 2 | 0 | 3 | 4 | 4 | 8 | 3
  ALTi, GRADE 0, GRADE 2: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  ALTi, GRADE 0, GRADE 3: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ALTi, GRADE 1, GRADE 0: number analyzed (Participants) | 4 | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 0
  ALTi, GRADE 1, GRADE 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 0
  ALTi, GRADE 1, GRADE 1: number analyzed (Participants) | 4 | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 0
  ALTi, GRADE 1, GRADE 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  ASTi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ASTi, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ASTi, GRADE 0, UNKNOWN: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ASTi, GRADE 0, GRADE 0: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 0 | 43 | 44 | 43 | 45 | 43 | 43 | 39 | 43 | 40 | 45
  ASTi, GRADE 0, GRADE 1: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 1 | 0 | 2 | 2 | 0 | 2 | 2 | 3 | 3 | 4 | 0
  ASTi, GRADE 0, GRADE 2: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  ASTi, GRADE 0, GRADE 4: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ASTi, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  ASTi, GRADE 1, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  ASTi, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ASTi, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  BUN, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  BUN, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  BUN, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  BUN, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 0 | 42 | 45 | 45 | 44 | 45 | 45 | 43 | 46 | 42 | 45
  BUN, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1
  BUN, GRADE 0, GRADE 2: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, GRADE 1, GRADE 0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 1, GRADE 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  CRE, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  CRE, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  CRE, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  CRE, GRADE 0, GRADE 0 | 44 | 46 | 45 | 46 | 46 | 46 | 43 | 47 | 45 | 46
  EOSi, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  EOSi, UNKNOWN, GRADE 0 | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 2 | 5 | 2
  EOSi, UNKNOWN, GRADE 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  EOSi, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  EOSi, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  EOSi, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, GRADE 0 | 43 | 40 | 39 | 44 | 45 | 44 | 40 | 43 | 36 | 43
  EOSi, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, GRADE 1 | 0 | 4 | 2 | 0 | 0 | 1 | 3 | 2 | 4 | 0
  EOSi, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  EOSi, GRADE 1, GRADE 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  EOSi, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  EOSi, GRADE 1, GRADE 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  HEMd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  HEMd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  HEMd, GRADE 0, GRADE 0: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 0 | 37 | 34 | 41 | 35 | 42 | 37 | 37 | 39 | 39 | 40
  HEMd, GRADE 0, GRADE 1: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 1 | 2 | 7 | 1 | 6 | 2 | 6 | 2 | 3 | 4 | 3
  HEMd, GRADE 0, GRADE 2: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  HEMd, GRADE 1, UNKNOWN: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  HEMd, GRADE 1, GRADE 0: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
  HEMd, GRADE 1, GRADE 1: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 1 | 2 | 1 | 1 | 3 | 0 | 1 | 2 | 0 | 0 | 0
  HEMd, GRADE 1, GRADE 2: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 2 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1
  HEMd, GRADE 2, GRADE 2: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0
  HEMd, GRADE 2, GRADE 2 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 0
  HEMd, GRADE 2, GRADE 3: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0
  HEMd, GRADE 2, GRADE 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
  HEMd, GRADE 3, GRADE 3: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  HEMd, GRADE 3, GRADE 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  LYMd, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  LYMd, UNKNOWN, GRADE 0 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  LYMd, UNKNOWN, GRADE 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  LYMd, UNKNOWN, GRADE 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  LYMd, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 0 | 41 | 41 | 39 | 44 | 40 | 44 | 43 | 41 | 38 | 40
  LYMd, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 1 | 2 | 1 | 0 | 1 | 3 | 1 | 0 | 4 | 1 | 4
  LYMd, GRADE 0, GRADE 2: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 0, GRADE 3: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 2: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NEUd, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 1
  NEUd, UNKNOWN, GRADE 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
  NEUd, UNKNOWN, GRADE 2: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  NEUd, UNKNOWN, GRADE 3: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  NEUd, GRADE 0, UNKNOWN: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  NEUd, GRADE 0, GRADE 0: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 0 | 37 | 35 | 40 | 36 | 37 | 39 | 37 | 35 | 36 | 37
  NEUd, GRADE 0, GRADE 1: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 1 | 4 | 4 | 1 | 4 | 2 | 4 | 2 | 4 | 2 | 3
  NEUd, GRADE 0, GRADE 2: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 2 | 0 | 1 | 0 | 2 | 1 | 1 | 3 | 1 | 1 | 1
  NEUd, GRADE 0, GRADE 3: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 3 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
  NEUd, GRADE 1, GRADE 0: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  NEUd, GRADE 1, GRADE 1: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
  NEUd, GRADE 1, GRADE 2: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
  NEUd, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 2, GRADE 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  NEUd, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  NEUd, GRADE 2, GRADE 2: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 2, GRADE 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  NEUd, GRADE 3, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NEUd, GRADE 3, GRADE 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  PLTCd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  PLTCd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  PLTCd, GRADE 0, UNKNOWN: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  PLTCd, GRADE 0, GRADE 0: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 0 | 42 | 45 | 44 | 43 | 46 | 45 | 43 | 45 | 44 | 45
  PLTCd, GRADE 0, GRADE 1: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  PLTCd, GRADE 0, GRADE 2: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  PLTCd, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 3: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  PLTCd, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  PLTCd, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  WBCd, UNKNOWN, GRADE 1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCd, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  WBCd, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WBCd, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, GRADE 0 | 41 | 43 | 44 | 41 | 41 | 46 | 42 | 42 | 40 | 41
  WBCd, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, GRADE 1 | 2 | 2 | 0 | 5 | 2 | 0 | 1 | 2 | 2 | 4
  WBCd, GRADE 0, GRADE 2: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, GRADE 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBCd, GRADE 1, GRADE 0: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0
  WBCd, GRADE 1, GRADE 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 0
  WBCd, GRADE 1, GRADE 1: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0
  WBCd, GRADE 1, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  WBCd, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBCd, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBCi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCi, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCi, GRADE 0, UNKNOWN: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WBCi, GRADE 0, GRADE 0: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 0 | 41 | 39 | 42 | 39 | 45 | 44 | 36 | 39 | 38 | 39
  WBCi, GRADE 0, GRADE 1: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 1 | 1 | 4 | 2 | 5 | 0 | 2 | 5 | 5 | 1 | 5
  WBCi, GRADE 0, GRADE 3: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCi, GRADE 1, GRADE 0: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
  WBCi, GRADE 1, GRADE 1: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 1 | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 2 | 2 | 1
  WBCi, GRADE 1, GRADE 2: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBCi, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCi, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

11. Primary Outcome: Number of Subjects With Change in Hematological and Biochemical Laboratory Results From Day 8 to Month 14+28 Days Versus Baseline by Toxicity Grading
Description: as for outcome 9
Time Frame: From Day 8 to Month 14 + 28 days
Population: Analysis was performed on the ES which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 45 | 46
Participants
  ALTi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALTi, GRADE 0, UNKNOWN: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALTi, GRADE 0, GRADE 0: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 0 | 38 | 38 | 39 | 42 | 40 | 41 | 38 | 39 | 30 | 40
  ALTi, GRADE 0, GRADE 1: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 1 | 1 | 8 | 3 | 2 | 4 | 3 | 5 | 4 | 13 | 6
  ALTi, GRADE 0, GRADE 2: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
  ALTi, GRADE 0, GRADE 3: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ALTi, GRADE 1, GRADE 0: number analyzed (Participants) | 4 | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 0
  ALTi, GRADE 1, GRADE 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 0
  ALTi, GRADE 1, GRADE 1: number analyzed (Participants) | 4 | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 0
  ALTi, GRADE 1, GRADE 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  ASTi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ASTi, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ASTi, UNKNOWN, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ASTi, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ASTi, GRADE 0, UNKNOWN: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ASTi, GRADE 0, GRADE 0: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 0 | 42 | 43 | 41 | 44 | 42 | 43 | 37 | 42 | 37 | 43
  ASTi, GRADE 0, GRADE 1: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 1 | 1 | 3 | 3 | 1 | 3 | 2 | 5 | 4 | 7 | 2
  ASTi, GRADE 0, GRADE 2: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  ASTi, GRADE 0, GRADE 4: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ASTi, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  ASTi, GRADE 1, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  ASTi, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ASTi, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  BUN, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  BUN, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  BUN, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  BUN, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 0 | 41 | 45 | 45 | 44 | 45 | 45 | 42 | 46 | 41 | 45
  BUN, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1
  BUN, GRADE 0, GRADE 2: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, GRADE 0, GRADE 3: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, GRADE 1, GRADE 0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 1, GRADE 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  CRE, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  CRE, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  CRE, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  CRE, GRADE 0, GRADE 0 | 44 | 46 | 45 | 46 | 46 | 46 | 43 | 47 | 45 | 46
  EOSi, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  EOSi, UNKNOWN, GRADE 0 | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 2 | 5 | 2
  EOSi, UNKNOWN, GRADE 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  EOSi, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  EOSi, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  EOSi, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, GRADE 0 | 42 | 40 | 39 | 43 | 45 | 44 | 39 | 42 | 34 | 43
  EOSi, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, GRADE 1 | 1 | 4 | 2 | 1 | 0 | 1 | 4 | 3 | 6 | 0
  EOSi, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  EOSi, GRADE 1, GRADE 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  EOSi, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  EOSi, GRADE 1, GRADE 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  HEMd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  HEMd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  HEMd, GRADE 0, GRADE 0: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 0 | 35 | 33 | 39 | 33 | 39 | 37 | 35 | 36 | 39 | 39
  HEMd, GRADE 0, GRADE 1: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 1 | 4 | 8 | 3 | 8 | 5 | 5 | 3 | 6 | 4 | 4
  HEMd, GRADE 0, GRADE 2: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  HEMd, GRADE 1, UNKNOWN: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  HEMd, GRADE 1, GRADE 0: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
  HEMd, GRADE 1, GRADE 1: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 1 | 2 | 1 | 1 | 3 | 0 | 1 | 2 | 0 | 0 | 0
  HEMd, GRADE 1, GRADE 2: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 2 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1
  HEMd, GRADE 1, GRADE 3: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HEMd, GRADE 2, GRADE 2: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0
  HEMd, GRADE 2, GRADE 2 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0
  HEMd, GRADE 2, GRADE 3: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0
  HEMd, GRADE 2, GRADE 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
  HEMd, GRADE 2, GRADE 4: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0
  HEMd, GRADE 2, GRADE 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HEMd, GRADE 3, GRADE 3: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  HEMd, GRADE 3, GRADE 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  LYMd, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  LYMd, UNKNOWN, GRADE 0 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 2 | 4 | 2
  LYMd, UNKNOWN, GRADE 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  LYMd, UNKNOWN, GRADE 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  LYMd, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  LYMd, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 0 | 40 | 41 | 39 | 44 | 40 | 44 | 43 | 38 | 38 | 40
  LYMd, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 1 | 3 | 1 | 0 | 1 | 3 | 1 | 0 | 7 | 1 | 4
  LYMd, GRADE 0, GRADE 2: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 0, GRADE 3: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 2: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NEUd, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 1
  NEUd, UNKNOWN, GRADE 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
  NEUd, UNKNOWN, GRADE 2: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  NEUd, UNKNOWN, GRADE 3: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  NEUd, GRADE 0, UNKNOWN: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  NEUd, GRADE 0, GRADE 0: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 0 | 36 | 34 | 37 | 35 | 36 | 38 | 34 | 35 | 34 | 34
  NEUd, GRADE 0, GRADE 1: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 1 | 5 | 4 | 2 | 5 | 3 | 5 | 5 | 4 | 4 | 6
  NEUd, GRADE 0, GRADE 2: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 2 | 0 | 2 | 2 | 2 | 1 | 1 | 3 | 1 | 1 | 1
  NEUd, GRADE 0, GRADE 3: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 3 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
  NEUd, GRADE 1, GRADE 0: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  NEUd, GRADE 1, GRADE 1: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  NEUd, GRADE 1, GRADE 2: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 2 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
  NEUd, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 2, GRADE 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  NEUd, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  NEUd, GRADE 2, GRADE 2: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 2, GRADE 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  NEUd, GRADE 3, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NEUd, GRADE 3, GRADE 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  PLTCd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  PLTCd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  PLTCd, GRADE 0, UNKNOWN: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  PLTCd, GRADE 0, GRADE 0: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 0 | 42 | 45 | 44 | 43 | 46 | 45 | 43 | 45 | 44 | 45
  PLTCd, GRADE 0, GRADE 1: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  PLTCd, GRADE 0, GRADE 2: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  PLTCd, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 3: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  PLTCd, GRADE 2, GRADE 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  PLTCd, GRADE 2, GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  WBCd, UNKNOWN, GRADE 1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCd, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  WBCd, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WBCd, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, GRADE 0 | 41 | 42 | 41 | 40 | 41 | 46 | 42 | 41 | 38 | 41
  WBCd, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, GRADE 1 | 2 | 3 | 3 | 6 | 2 | 0 | 1 | 3 | 4 | 4
  WBCd, GRADE 0, GRADE 2: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, GRADE 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBCd, GRADE 1, GRADE 0: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0
  WBCd, GRADE 1, GRADE 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 0
  WBCd, GRADE 1, GRADE 1: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0
  WBCd, GRADE 1, GRADE 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  WBCd, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBCd, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBCi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCi, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCi, GRADE 0, UNKNOWN: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WBCi, GRADE 0, GRADE 0: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 0 | 39 | 39 | 40 | 37 | 43 | 43 | 35 | 37 | 36 | 36
  WBCi, GRADE 0, GRADE 1: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 1 | 3 | 4 | 4 | 6 | 2 | 3 | 5 | 6 | 3 | 7
  WBCi, GRADE 0, GRADE 2: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
  WBCi, GRADE 0, GRADE 3: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCi, GRADE 1, GRADE 0: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
  WBCi, GRADE 1, GRADE 1: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 1 | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 1
  WBCi, GRADE 1, GRADE 2: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCi, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCi, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

12. Primary Outcome: Number of Subjects With Change in Hematological and Biochemical Laboratory Results From Day 8 to Month 26 Versus Baseline by Toxicity Grading
Description: as for outcome 9
Time Frame: From Day 8 to Month 26
Population: Analysis was performed on the ES which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 45 | 46
Participants
  ALTi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ALTi, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALTi, GRADE 0, UNKNOWN: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALTi, GRADE 0, GRADE 0: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 0 | 38 | 38 | 39 | 42 | 40 | 39 | 37 | 38 | 29 | 40
  ALTi, GRADE 0, GRADE 1: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 1 | 1 | 8 | 3 | 2 | 4 | 5 | 6 | 5 | 14 | 6
  ALTi, GRADE 0, GRADE 2: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
  ALTi, GRADE 0, GRADE 3: number analyzed (Participants) | 40 | 46 | 43 | 45 | 45 | 45 | 44 | 44 | 43 | 46
  ALTi, GRADE 0, GRADE 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ALTi, GRADE 1, GRADE 0: number analyzed (Participants) | 4 | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 0
  ALTi, GRADE 1, GRADE 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 0
  ALTi, GRADE 1, GRADE 1: number analyzed (Participants) | 4 | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 0
  ALTi, GRADE 1, GRADE 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
  ASTi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ASTi, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ASTi, UNKNOWN, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ASTi, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ASTi, GRADE 0, UNKNOWN: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ASTi, GRADE 0, GRADE 0: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 0 | 42 | 42 | 41 | 44 | 42 | 42 | 36 | 42 | 37 | 43
  ASTi, GRADE 0, GRADE 1: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 1 | 1 | 4 | 3 | 1 | 3 | 1 | 6 | 4 | 7 | 2
  ASTi, GRADE 0, GRADE 2: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 2 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 1
  ASTi, GRADE 0, GRADE 4: number analyzed (Participants) | 44 | 46 | 45 | 46 | 46 | 45 | 43 | 46 | 45 | 46
  ASTi, GRADE 0, GRADE 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ASTi, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  ASTi, GRADE 1, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  ASTi, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ASTi, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  BUN, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  BUN, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  BUN, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  BUN, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 0 | 40 | 45 | 45 | 44 | 45 | 45 | 42 | 46 | 41 | 45
  BUN, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 1 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1
  BUN, GRADE 0, GRADE 2: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, GRADE 0, GRADE 3: number analyzed (Participants) | 43 | 46 | 45 | 46 | 46 | 46 | 44 | 47 | 43 | 46
  BUN, GRADE 0, GRADE 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, GRADE 1, GRADE 0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 1, GRADE 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, GRADE 1, GRADE 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 1, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BUN, GRADE 2, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  CRE, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  CRE, UNKNOWN, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  CRE, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  CRE, GRADE 0, GRADE 0 | 44 | 46 | 45 | 46 | 46 | 46 | 43 | 47 | 45 | 46
  EOSi, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  EOSi, UNKNOWN, GRADE 0 | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 2 | 5 | 2
  EOSi, UNKNOWN, GRADE 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  EOSi, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  EOSi, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  EOSi, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, GRADE 0 | 42 | 40 | 39 | 43 | 45 | 44 | 38 | 41 | 34 | 42
  EOSi, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 44 | 41 | 44 | 45 | 45 | 44 | 45 | 40 | 43
  EOSi, GRADE 0, GRADE 1 | 1 | 4 | 2 | 1 | 0 | 1 | 5 | 4 | 6 | 1
  EOSi, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  EOSi, GRADE 1, GRADE 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  EOSi, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  EOSi, GRADE 1, GRADE 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  HEMd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  HEMd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  HEMd, GRADE 0, GRADE 0: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 0 | 33 | 32 | 37 | 31 | 38 | 36 | 35 | 35 | 37 | 39
  HEMd, GRADE 0, GRADE 1: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 1 | 5 | 9 | 5 | 7 | 6 | 6 | 3 | 6 | 5 | 4
  HEMd, GRADE 0, GRADE 2: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 2 | 1 | 0 | 0 | 4 | 0 | 1 | 1 | 1 | 0 | 0
  HEMd, GRADE 0, GRADE 3: number analyzed (Participants) | 39 | 41 | 42 | 42 | 44 | 43 | 39 | 42 | 43 | 43
  HEMd, GRADE 0, GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  HEMd, GRADE 1, UNKNOWN: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  HEMd, GRADE 1, GRADE 0: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
  HEMd, GRADE 1, GRADE 1: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 1 | 2 | 1 | 1 | 3 | 0 | 1 | 2 | 0 | 0 | 0
  HEMd, GRADE 1, GRADE 2: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 2 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1
  HEMd, GRADE 1, GRADE 3: number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 2 | 4 | 2 | 1 | 2
  HEMd, GRADE 1, GRADE 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HEMd, GRADE 2, GRADE 2: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0
  HEMd, GRADE 2, GRADE 2 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0
  HEMd, GRADE 2, GRADE 3: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0
  HEMd, GRADE 2, GRADE 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
  HEMd, GRADE 2, GRADE 4: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0
  HEMd, GRADE 2, GRADE 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HEMd, GRADE 3, GRADE 3: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  HEMd, GRADE 3, GRADE 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  LYMd, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  LYMd, UNKNOWN, GRADE 0 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 2 | 4 | 2
  LYMd, UNKNOWN, GRADE 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  LYMd, UNKNOWN, GRADE 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  LYMd, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  LYMd, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 0 | 39 | 40 | 39 | 44 | 40 | 44 | 43 | 37 | 38 | 40
  LYMd, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 1 | 4 | 1 | 0 | 1 | 3 | 1 | 0 | 8 | 1 | 4
  LYMd, GRADE 0, GRADE 2: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 2 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 0, GRADE 3: number analyzed (Participants) | 43 | 45 | 39 | 45 | 44 | 45 | 44 | 45 | 39 | 44
  LYMd, GRADE 0, GRADE 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 1, GRADE 1: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 2: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  LYMd, GRADE 1, GRADE 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  LYMd, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NEUd, UNKNOWN, GRADE 0: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 1
  NEUd, UNKNOWN, GRADE 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
  NEUd, UNKNOWN, GRADE 2: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  NEUd, UNKNOWN, GRADE 3: number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 5 | 2
  NEUd, UNKNOWN, GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  NEUd, GRADE 0, UNKNOWN: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  NEUd, GRADE 0, GRADE 0: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 0 | 35 | 34 | 37 | 35 | 36 | 36 | 34 | 35 | 34 | 34
  NEUd, GRADE 0, GRADE 1: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 1 | 5 | 4 | 2 | 5 | 3 | 6 | 5 | 4 | 4 | 6
  NEUd, GRADE 0, GRADE 2: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 2 | 1 | 2 | 2 | 2 | 1 | 2 | 3 | 1 | 1 | 1
  NEUd, GRADE 0, GRADE 3: number analyzed (Participants) | 41 | 41 | 41 | 44 | 41 | 44 | 43 | 41 | 39 | 41
  NEUd, GRADE 0, GRADE 3 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
  NEUd, GRADE 1, GRADE 0: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  NEUd, GRADE 1, GRADE 1: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  NEUd, GRADE 1, GRADE 2: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1
  NEUd, GRADE 1, GRADE 2 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
  NEUd, GRADE 2, GRADE 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 2, GRADE 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  NEUd, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  NEUd, GRADE 2, GRADE 2: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2
  NEUd, GRADE 2, GRADE 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  NEUd, GRADE 3, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NEUd, GRADE 3, GRADE 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  PLTCd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  PLTCd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  PLTCd, GRADE 0, UNKNOWN: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  PLTCd, GRADE 0, GRADE 0: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 0 | 42 | 45 | 44 | 43 | 46 | 44 | 43 | 45 | 44 | 45
  PLTCd, GRADE 0, GRADE 1: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  PLTCd, GRADE 0, GRADE 2: number analyzed (Participants) | 44 | 45 | 45 | 44 | 46 | 46 | 44 | 46 | 44 | 45
  PLTCd, GRADE 0, GRADE 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  PLTCd, GRADE 1, GRADE 0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 3: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  PLTCd, GRADE 1, GRADE 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  PLTCd, GRADE 2, GRADE 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  PLTCd, GRADE 2, GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCd, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCd, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  WBCd, UNKNOWN, GRADE 1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCd, UNKNOWN, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  WBCd, GRADE 0, UNKNOWN: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WBCd, GRADE 0, GRADE 0: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, GRADE 0 | 39 | 42 | 41 | 40 | 41 | 46 | 42 | 41 | 38 | 41
  WBCd, GRADE 0, GRADE 1: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, GRADE 1 | 4 | 3 | 3 | 6 | 2 | 0 | 1 | 3 | 4 | 4
  WBCd, GRADE 0, GRADE 2: number analyzed (Participants) | 43 | 45 | 44 | 46 | 44 | 46 | 44 | 44 | 42 | 45
  WBCd, GRADE 0, GRADE 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBCd, GRADE 1, GRADE 0: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0
  WBCd, GRADE 1, GRADE 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0
  WBCd, GRADE 1, GRADE 1: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 0
  WBCd, GRADE 1, GRADE 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  WBCd, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBCd, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBCi, UNKNOWN, GRADE 0: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCi, UNKNOWN, GRADE 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  WBCi, GRADE 0, UNKNOWN: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  WBCi, GRADE 0, GRADE 0: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 0 | 37 | 38 | 40 | 37 | 43 | 43 | 35 | 37 | 36 | 36
  WBCi, GRADE 0, GRADE 1: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 1 | 5 | 5 | 4 | 6 | 2 | 3 | 5 | 6 | 3 | 7
  WBCi, GRADE 0, GRADE 2: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
  WBCi, GRADE 0, GRADE 3: number analyzed (Participants) | 42 | 43 | 44 | 44 | 45 | 46 | 42 | 44 | 40 | 44
  WBCi, GRADE 0, GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCi, GRADE 1, GRADE 0: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
  WBCi, GRADE 1, GRADE 1: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 1 | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 1
  WBCi, GRADE 1, GRADE 2: number analyzed (Participants) | 2 | 2 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 1
  WBCi, GRADE 1, GRADE 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCi, GRADE 2, GRADE 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBCi, GRADE 2, GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

13. Primary Outcome: Number of Subjects With Any Medically-attended Adverse Events (MAEs)
Description: MAEs are defined as events for which the subject receives medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination.
Time Frame: During the entire study period (from Day 1 up to Month 26)
Population: Analysis was performed on the ES which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 45 | 46 | 47 | 47 | 48 | 47 | 47 | 48 | 46 | 47
Participants | 21 | 16 | 20 | 23 | 21 | 14 | 19 | 18 | 23 | 20

14. Primary Outcome: Number of Subjects Reporting Any Potential Immune-mediated Diseases (pIMDs)
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: During the entire study period (from Day 1 up to Month 26)
Population: Analysis was performed on the ES which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 45 | 46 | 47 | 47 | 48 | 47 | 47 | 48 | 46 | 47
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

15. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: SAEs include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 1 up to Month 26)
Population: Analysis was performed on the ES which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 45 | 46 | 47 | 47 | 48 | 47 | 47 | 48 | 46 | 47
Participants | 2 | 1 | 1 | 2 | 2 | 2 | 0 | 2 | 2 | 3

16. Primary Outcome: Number of Seropositive Subjects for Anti-H1 Stalk Antibodies Measured by Enzyme-linked Immunosorbent Assay (ELISA)- Day 1
Description: Anti-H1 stalk immune response measured by ELISA. A seropositive subject is a subject whose concentration is greater than or equal to the cut-off value: ELISA cut-off = 66 ELISA.Unit per milliliter (EL.U/mL).
Time Frame: At Day 1
Population: Analysis of immunogenicity was performed on the Per-Protocol Set (PPS) which included all eligible subjects according to protocol and for whom immunogenicity results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 45 | 46 | 47 | 47 | 48 | 47 | 47 | 46 | 44 | 45
Participants | 45 | 46 | 47 | 47 | 48 | 47 | 47 | 46 | 44 | 45

17. Primary Outcome: Number of Seropositive Subjects for Anti-H1 Stalk Antibodies Measured by ELISA- Day 29
Description: Anti-H1 stalk immune response measured by ELISA. A seropositive subject is a subject whose concentration is greater than or equal to the cut-off value: ELISA cut-off = 66 EL.U/mL.
Time Frame: At Day 29
Population: Analysis of immunogenicity was performed on the PPS which included all eligible subjects according to protocol and for whom immunogenicity results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
Participants | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40

18. Primary Outcome: Number of Seropositive Subjects for Anti-H1 Stalk Antibodies Measured by ELISA- Day 85
Description: as for outcome 17
Time Frame: At Day 85
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
Participants | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38

19. Primary Outcome: Concentrations of Serum H1 Stalk Antibodies Measured by ELISA- Day 1
Description: Concentrations are presented as Geometric Mean Concentrations (GMCs) and measured by ELISA. ELISA cut-off = 66 EL.U/mL.
Time Frame: At Day 1
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 45 | 46 | 47 | 47 | 48 | 47 | 47 | 46 | 44 | 45
EL.U/mL | 8887.9 [7004.9 to 11277.1] | 8719.3 [6547.0 to 11612.3] | 9691 [7593.7 to 12367.7] | 9121 [7180.0 to 11586.6] | 9948.6 [8106.2 to 12209.8] | 8555.5 [6980.1 to 10486.4] | 9019.6 [7263.5 to 11200.2] | 9278.2 [7430.7 to 11585.1] | 9039.3 [6930.7 to 11789.5] | 9160 [7225.7 to 11612.2]

20. Primary Outcome: Concentrations of Serum H1 Stalk Antibodies Measured by ELISA- Day 29
Description: Concentrations are presented as GMCs and measured by ELISA. ELISA cut-off = 66 EL.U/mL.
Time Frame: At Day 29
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
EL.U/mL | 112973.2 [90888.2 to 140424.5] | 45645 [35289.4 to 59039.5] | 116596.8 [93869.6 to 144826.6] | 61634.2 [49810.3 to 76264.7] | 46596.2 [38306.7 to 56679.5] | 67114.6 [54649.7 to 82422.6] | 35580.2 [24654.2 to 51348.2] | 20398.6 [16362.4 to 25430.5] | 36426.2 [29124.8 to 45558.0] | 21938.1 [18037.8 to 26681.8]

21. Primary Outcome: Concentrations of Serum H1 Stalk Antibodies Measured by ELISA- Day 85
Description: Concentrations are presented as GMCs and measured by ELISA. ELISA cut-off = 66 EL.U/mL.
Time Frame: At Day 85
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
EL.U/mL | 45351.6 [36766.7 to 55941.1] | 28437.5 [21623.4 to 37398.9] | 74639.7 [59986.3 to 92872.6] | 30419.3 [23619.9 to 39176.0] | 25718.6 [20748.8 to 31878.8] | 48775.9 [40697.7 to 58457.7] | 28617.8 [19448.1 to 42110.9] | 15105.9 [12007.7 to 19003.6] | 37911.4 [30149.4 to 47671.7] | 16749.9 [13471.8 to 20825.8]

22. Primary Outcome: Number of Seropositive Subjects for Anti-H1 Stalk Antibodies Measured by Microneutralization (MN) Assay - Day 1
Description: Anti-H1 stalk immune response measured by MN are expressed in 1/DILUTION (DIL). The functionality of the stalk-reactive antibodies is evaluated by MN assays developed using chimeric viruses. A seropositive subject is a subject whose titer is greater than or equal to the cut-off value: MN cut-off = 20 1/DIL.
Time Frame: At Day 1
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 44 | 44 | 45 | 46 | 44 | 46 | 45 | 43 | 42 | 41
Participants | 32 | 34 | 35 | 36 | 33 | 40 | 37 | 34 | 31 | 33

23. Primary Outcome: Number of Seropositive Subjects for Anti-H1 Stalk Antibodies Measured by MN Assay - Day 29
Description: Anti-H1 stalk immune response measured by MN are expressed in 1/DIL. The functionality of the stalk-reactive antibodies is evaluated by MN assays developed using chimeric viruses. A seropositive subject is a subject whose titer is greater than or equal to the cut-off value: MN cut-off = 20 1/DIL.
Time Frame: At Day 29
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 40 | 40 | 41 | 42 | 37 | 41 | 39 | 40
Participants | 43 | 40 | 40 | 40 | 41 | 41 | 36 | 41 | 37 | 40

24. Primary Outcome: Number of Seropositive Subjects for Anti-H1 Stalk Antibodies Measured by MN Assay - Day 85
Description: as for outcome 23
Time Frame: At Day 85
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 38 | 36 | 34 | 33 | 39 | 35 | 34 | 34 | 35 | 38
Participants | 36 | 35 | 34 | 31 | 38 | 35 | 30 | 32 | 35 | 37

25. Primary Outcome: Titers for Serum H1 Stalk Antibodies Measured by MN Assay - Day 1
Description: Titers are presented as GMTs and measured by MN assay. MN cut-off = 20 1/DIL.
Time Frame: At Day 1
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 44 | 44 | 45 | 46 | 44 | 46 | 45 | 43 | 42 | 41
Titer | 40.6 [29.4 to 56.1] | 45.4 [33.4 to 61.6] | 45.9 [34.2 to 61.8] | 45.8 [34.5 to 60.8] | 41.9 [30.7 to 57.3] | 45.1 [35.0 to 58.2] | 44.6 [34.4 to 57.7] | 43.4 [32.4 to 58.0] | 42.7 [31.2 to 58.6] | 38 [28.8 to 50.2]

26. Primary Outcome: Titers for Serum H1 Stalk Antibodies Measured by MN Assay - Day 29
Description: Titers are presented as GMTs and measured by MN assay. MN cut-off = 20 1/DIL.
Time Frame: At Day 29
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 40 | 40 | 41 | 42 | 37 | 41 | 39 | 40
Titer | 100.3 [88.1 to 114.1] | 109.3 [94.0 to 127.0] | 113.1 [96.5 to 132.6] | 105.6 [91.0 to 122.5] | 96.4 [83.2 to 111.6] | 89.8 [73.0 to 110.5] | 86.2 [69.9 to 106.3] | 80 [66.6 to 96.1] | 74.5 [59.6 to 93.2] | 87.2 [75.6 to 100.7]

27. Primary Outcome: Titers for Serum H1 Stalk Antibodies Measured by MN Assay - Day 85
Description: Titers are presented as GMTs and measured by MN assay. MN cut-off = 20 1/DIL.
Time Frame: At Day 85
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 38 | 36 | 34 | 33 | 39 | 35 | 34 | 34 | 35 | 38
Titer | 73 [58.3 to 91.5] | 98.9 [81.5 to 119.9] | 122.7 [108.9 to 138.3] | 59.6 [45.9 to 77.4] | 87.4 [71.1 to 107.6] | 109.8 [93.0 to 129.8] | 55.4 [41.3 to 74.3] | 75.3 [56.4 to 100.4] | 88.3 [74.2 to 105.2] | 86.1 [70.2 to 105.5]

28. Primary Outcome: Percentage of Subjects With a ≥ 4-fold Increase of Anti-H1 Stalk Antibody Concentration Measured by ELISA - Day 29
Description: Percentage of subjects with an equal or greater than (≥) 4-fold increase of anti-H1 stalk antibody concentration, from Day 1, is calculated with exact 95% CI by ELISA.
Time Frame: At Day 29, compared to pre-vaccination at Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
Percentage of subjects | 88.4 [74.9 to 96.1] | 60 [43.3 to 75.1] | 87.8 [73.8 to 95.9] | 70 [53.5 to 83.4] | 52.4 [36.4 to 68.0] | 83.3 [68.6 to 93.0] | 35.1 [20.2 to 52.5] | 24.4 [12.4 to 40.3] | 38.5 [23.4 to 55.4] | 15 [5.7 to 29.8]

29. Primary Outcome: Percentage of Subjects With a ≥ 4-fold Increase of Anti-H1 Stalk Antibody Concentration Measured by ELISA - Day 85
Description: Percentage of subjects with a ≥ 4-fold increase of anti-H1 stalk antibody concentration, from Day 1, is calculated with exact 95% CI by ELISA.
Time Frame: At Day 85, compared to pre-vaccination at Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
Percentage of subjects | 51.3 [34.8 to 67.6] | 44.4 [27.9 to 61.9] | 79.4 [62.1 to 91.3] | 37.1 [21.5 to 55.1] | 20.5 [9.3 to 36.5] | 80 [63.1 to 91.6] | 29.4 [15.1 to 47.5] | 8.8 [1.9 to 23.7] | 37.1 [21.5 to 55.1] | 7.9 [1.7 to 21.4]

30. Primary Outcome: Percentage of Subjects With a ≥ 4-fold Increase of Anti-H1 Stalk Titer Measured by MN Assay - Day 29
Description: Percentage of subjects with a ≥ 4-fold increase of anti-H1 stalk antibody titer from Day 1, is calculated with exact 95% CI by MN assay.
Time Frame: At Day 29, compared to pre-vaccination at Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 42 | 38 | 38 | 39 | 38 | 41 | 35 | 38 | 37 | 36
Percentage of subjects | 40.5 [25.6 to 56.7] | 39.5 [24.0 to 56.6] | 31.6 [17.5 to 48.7] | 41 [25.6 to 57.9] | 36.8 [21.8 to 54.0] | 31.7 [18.1 to 48.1] | 34.3 [19.1 to 52.2] | 26.3 [13.4 to 43.1] | 29.7 [15.9 to 47.0] | 36.1 [20.8 to 53.8]

31. Primary Outcome: Percentage of Subjects With a ≥ 4-fold Increase of Anti-H1 Stalk Titer Measured by MN Assay - Day 85
Description: as for outcome 30
Time Frame: At Day 85, compared to pre-vaccination at Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 37 | 34 | 32 | 33 | 35 | 34 | 33 | 32 | 33 | 34
Percentage of subjects | 29.7 [15.9 to 47.0] | 38.2 [22.2 to 56.4] | 34.4 [18.6 to 53.2] | 15.2 [5.1 to 31.9] | 31.4 [16.9 to 49.3] | 41.2 [24.6 to 59.3] | 21.2 [9.0 to 38.9] | 18.8 [7.2 to 36.4] | 33.3 [18.0 to 51.8] | 41.2 [24.6 to 59.3]

32. Primary Outcome: Percentage of Subjects With a ≥ 10-fold Increase of Anti-H1 Stalk Antibody Concentration Measured by ELISA - Day 29
Description: Percentage of subjects with a ≥ 10-fold increase of anti-H1 stalk antibody concentration, from Day 1, is calculated with exact 95% CI by ELISA.
Time Frame: At Day 29, compared to pre-vaccination at Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
Percentage of subjects | 58.1 [42.1 to 73.0] | 35 [20.6 to 51.7] | 61 [44.5 to 75.8] | 30 [16.6 to 46.5] | 21.4 [10.3 to 36.8] | 42.9 [27.7 to 59.0] | 13.5 [4.5 to 28.8] | 2.4 [0.1 to 12.9] | 15.4 [5.9 to 30.5] | 2.5 [0.1 to 13.2]

33. Primary Outcome: Percentage of Subjects With a ≥ 10-fold Increase of Anti-H1 Stalk Antibody Concentration Measured by ELISA - Day 85
Description: as for outcome 32
Time Frame: At Day 85, compared to pre-vaccination at Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
Percentage of subjects | 12.8 [4.3 to 27.4] | 5.6 [0.7 to 18.7] | 47.1 [29.8 to 64.9] | 17.1 [6.6 to 33.6] | 5.1 [0.6 to 17.3] | 25.7 [12.5 to 43.3] | 17.6 [6.8 to 34.5] | 2.9 [0.1 to 15.3] | 14.3 [4.8 to 30.3] | 5.3 [0.6 to 17.7]

34. Primary Outcome: Percentage of Subjects With a ≥ 10-fold Increase of Anti-H1 Stalk Titer Measured by MN Assay - Day 29
Description: Percentage of subjects with a ≥ 10-fold increase of anti-H1 stalk antibody titer from Day 1, is calculated with exact 95% CI by MN assay.
Time Frame: At Day 29, compared to pre-vaccination at Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 42 | 38 | 38 | 39 | 38 | 41 | 35 | 38 | 37 | 36
Percentage of subjects | 7.1 [1.5 to 19.5] | 7.9 [1.7 to 21.4] | 10.5 [2.9 to 24.8] | 5.1 [0.6 to 17.3] | 7.9 [1.7 to 21.4] | 4.9 [0.6 to 16.5] | 8.6 [1.8 to 23.1] | 2.6 [0.1 to 13.8] | 2.7 [0.1 to 14.2] | 2.8 [0.1 to 14.5]

35. Primary Outcome: Percentage of Subjects With a ≥ 10-fold Increase of Anti-H1 Stalk Titer Measured by MN Assay - Day 85
Description: as for outcome 34
Time Frame: At Day 85, compared to pre-vaccination at Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 37 | 34 | 32 | 33 | 35 | 34 | 33 | 32 | 33 | 34
Percentage of subjects | 2.7 [0.1 to 14.2] | 8.8 [1.9 to 23.7] | 15.6 [5.3 to 32.8] | 3 [0.1 to 15.8] | 8.6 [1.8 to 23.1] | 8.8 [1.9 to 23.7] | 0 [0.0 to 10.6] | 6.3 [0.8 to 20.8] | 3 [0.1 to 15.8] | 2.9 [0.1 to 15.3]

36. Primary Outcome: Mean Geometric Increase (MGI) for Anti-H1 Stalk Antibody Concentration Measured by ELISA - Day 29
Description: MGI is defined as the geometric mean of the fold increase in serum HI concentration post-vaccination compared to Day 1
Time Frame: At Day 29, compared to pre-vaccination at Day 1
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
Ratio | 12.4 [9.2 to 16.7] | 5.9 [4.4 to 8.0] | 12.6 [9.2 to 17.1] | 6.8 [4.9 to 9.5] | 4.7 [3.6 to 6.2] | 8.1 [6.2 to 10.5] | 4.2 [2.9 to 6.2] | 2.3 [1.8 to 3.0] | 3.9 [2.8 to 5.4] | 2.4 [1.9 to 2.9]

37. Primary Outcome: MGI for Anti-H1 Stalk Antibody Concentration Measured by ELISA - Day 85
Description: MGI is defined as the geometric mean of the fold increase in serum HI concentration post-vaccination compared to Day 1
Time Frame: At Day 85, compared to pre-vaccination at Day 1
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
Ratio | 5 [3.9 to 6.5] | 3.4 [2.6 to 4.5] | 8.1 [6.1 to 10.8] | 3.4 [2.4 to 4.9] | 2.6 [2.1 to 3.2] | 6.3 [5.0 to 7.9] | 3.4 [2.3 to 5.0] | 1.7 [1.4 to 2.1] | 3.8 [2.7 to 5.5] | 1.8 [1.5 to 2.3]

38. Primary Outcome: MGI for Anti-H1 Stalk Antibody Titer Measured by MN Assay - Day 29
Description: MGI is defined as the geometric mean of the fold increase in serum HI titer post-vaccination compared to Day 1
Time Frame: At Day 29, compared to pre-vaccination at Day 1
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 42 | 38 | 38 | 39 | 38 | 41 | 35 | 38 | 37 | 36
Ratio | 2.4 [1.7 to 3.3] | 2.6 [1.9 to 3.6] | 2.4 [1.8 to 3.3] | 2.3 [1.7 to 3.2] | 2.3 [1.7 to 3.2] | 2 [1.5 to 2.7] | 2.3 [1.7 to 3.2] | 1.9 [1.4 to 2.5] | 1.7 [1.2 to 2.4] | 2.2 [1.6 to 3.1]

39. Primary Outcome: MGI for Anti-H1 Stalk Antibody Titer Measured by MN Assay - Day 85
Description: MGI is defined as the geometric mean of the fold increase in serum HI titer post-vaccination compared to Day 1
Time Frame: At Day 85, compared to pre-vaccination at Day 1
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 37 | 34 | 32 | 33 | 35 | 34 | 33 | 32 | 33 | 34
Ratio | 1.6 [1.2 to 2.2] | 2.2 [1.5 to 3.2] | 2.5 [1.7 to 3.7] | 1.1 [0.8 to 1.6] | 2 [1.5 to 2.8] | 2.5 [1.7 to 3.5] | 1.2 [0.9 to 1.7] | 1.6 [1.1 to 2.2] | 2 [1.4 to 2.8] | 2.4 [1.7 to 3.3]

40. Secondary Outcome: Adjusted GMCs for Anti-H1 HA Stalk Antibody Measured by ELISA
Description: The adjusted GMCs are presented to evaluate the adjuvant effect post-dose 1 and post-dose 2.
Time Frame: 28 days post priming dose(s) i.e. at Day 29 for 1 priming dose groups and at Day 85 for 2 priming doses groups
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 34 | 40 | 42 | 35 | 37 | 41 | 35 | 40
EL.U/mL | 112206.4 [91362.2 to 137806.3] | 47432.6 [38317.4 to 58716.2] | 73945.6 [58686.6 to 93172.2] | 61356.7 [49582.3 to 75927] | 45346.6 [36827 to 55837.2] | 50602.8 [40283.4 to 63565.8] | 36159.3 [28972.3 to 45129] | 20403.5 [16531.4 to 25182.7] | 36826.9 [29320 to 46255.8] | 21675.2 [17515.2 to 26823.1]
Statistical Analysis 1: Comparison: D-SUIV Adjuvanted Group 1 vs D-SUIV Unadjuvanted Group 1; To evaluate the adjuvant effect of AS03 (Pooling of results at Day 29 of D-SUIV Adjuvant Group 1, at Day 29 of D-SUIV Adjuvant Group 2 and Day 85 of D-SUIV Adjuvant Group 3) on the humoral immune response for anti-H1 stalk antibody by ELISA at Day 29 and Day 85 (i.e. 28 days post-vaccination) when compared to the non-adjuvanted formulations (Pooling of results at Day 29 of D-SUIV Unadjuvanted Group 1, at Day 29 of D-SUIV Unadjuvanted Group 2 and Day 85 of D-SUIV Unadjuvanted Group 3); Test type: Equivalence — The use of the adjuvant (AS03) is to be considered justified if the lower limit of the 94.46% CI of the GMC ratio (adjuvanted vs non-adjuvanted) is > 1.50; Dunnett's t test; Comparison performed using a 2-sided alpha=0.1 and Dunnett adjustment for multiple comparisons,; GMC ratio = 2.47, 94.46% CI 2-sided [2.06 to 2.95]
Statistical Analysis 2: Comparison: D-SUIV Adjuvanted Group 4 vs D-SUIV Unadjuvanted Group 1; To evaluate the adjuvant effect of AS01 (Pooling of results at Day 29 of D-SUIV Adjuvant Group 4, at Day 29 of D-SUIV Adjuvant Group 5 and Day 85 of D-SUIV Adjuvant Group 6) on the humoral immune response for anti-H1 stalk antibody by ELISA at Day 29 and Day 85 (i.e. 28 days post-vaccination) when compared to the non-adjuvanted formulations (Pooling of results at Day 29 of D-SUIV Unadjuvanted Group 1, at Day 29 of D-SUIV Unadjuvanted Group 2 and Day 85 of D-SUIV Unadjuvanted Group 3); Test type: Equivalence — The use of the adjuvant (AS01) is to be considered justified if the lower limit of the 94.46% CI of the GMC ratio (adjuvanted vs non-adjuvanted) is > 1.50; Dunnett's t test; Comparison performed using a 2-sided alpha=0.1 and Dunnett adjustment for multiple comparisons,; GMC ratio = 1.75, 94.46% CI 2-sided [1.46 to 2.1]

41. Secondary Outcome: Concentrations of Serum H1 Stalk Antibodies Measured by ELISA- Month 8 to 26
Description: Concentrations are presented as GMCs and measured by ELISA. ELISA cut-off = 66 EL.U/mL.
Time Frame: At Month 8, Month 14, Month 14 + 28 days, Month 20 and Month 26.
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
EL.U/mL
  M8 | 27068.3 [21884.3 to 33480.4] | 17155.9 [13158.7 to 22367.4] | 41759.7 [32814.0 to 53144.1] | 18915.3 [15026.4 to 23810.7] | 15092.4 [12226.1 to 18630.8] | 25279.1 [20711.4 to 30854.2] | 19028.4 [13706.8 to 26416.0] | 11024.8 [8751.5 to 13888.6] | 22359.8 [18089.1 to 27638.8] | 13142.1 [10306.0 to 16758.7]
  M14: number analyzed (Participants) | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  M14 | 22687.1 [18078.5 to 28470.4] | 17662.4 [14339.6 to 21755.1] | 37282.2 [29437.7 to 47216.9] | 20146.8 [15305.9 to 26518.8] | 16645.4 [12389.7 to 22362.8] | 24615 [19677.5 to 30791.4] | 16969.8 [11848.5 to 24304.6] | 10820.3 [8524.9 to 13733.9] | 22791.5 [17767.3 to 29236.4] | 12458.4 [9721.6 to 15965.7]
  M14+28 days: number analyzed (Participants) | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  M14+28 days | 49594 [39888.4 to 61661.1] | 92885.6 [73985.7 to 116613.7] | 73078 [62288.9 to 85736.0] | 36709.7 [30186.1 to 44643.2] | 75155.7 [56729.2 to 99567.4] | 52026.4 [42254.7 to 64057.8] | 22653.6 [16071.5 to 31931.4] | 29508.2 [21062.2 to 41341.1] | 38364 [30403.9 to 48408.1] | 17593.3 [13932.1 to 22216.6]
  M20: number analyzed (Participants) | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  M20 | 27648.6 [22712.3 to 33657.7] | 36133.6 [29063.7 to 44923.2] | 38120.3 [30433.7 to 47748.2] | 21916.1 [17219.1 to 27894.4] | 31396.4 [24953.9 to 39502.2] | 29988.8 [24033.9 to 37419.1] | 18408.1 [12608.3 to 26875.7] | 16632.9 [12484.8 to 22159.2] | 23145.3 [18447.2 to 29039.9] | 12635.2 [9489.2 to 16824.1]
  M26: number analyzed (Participants) | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  M26 | 22850.2 [18790.0 to 27787.8] | 29027.2 [23343.2 to 36095.3] | 32635.4 [26013.9 to 40942.3] | 18266 [14093.9 to 23673.1] | 27491.3 [20448.3 to 36960.2] | 25059.4 [19893.4 to 31567.0] | 18220.9 [12067.9 to 27511.0] | 14269 [10104.9 to 20149.0] | 21673.7 [17482.9 to 26869.2] | 12050.6 [8943.4 to 16237.5]

42. Secondary Outcome: Number of Seropositive Subjects for Anti-H1 Stalk Antibodies Measured by ELISA- Month 8 to 26
Description: as for outcome 17
Time Frame: At Month 8, Month 14, Month 14 + 28 days, Month 20 and Month 26.
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
Participants
  M8 | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
  M14: number analyzed (Participants) | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  M14 | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  M14+28 days: number analyzed (Participants) | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  M14+28 days | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  M20: number analyzed (Participants) | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  M20 | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  M26: number analyzed (Participants) | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  M26 | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23

43. Secondary Outcome: Percentage of Subjects With a ≥ 4-fold Increase of Anti-H1 Stalk Antibody Concentration, Measured by ELISA - Month 8 to 26.
Description: as for outcome 29
Time Frame: At Month 8, Month 14, Month 14 + 28 days, Month 20 and Month 26, compared to Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
Percentage of subjects
  M8 | 23.1 [11.1 to 39.3] | 23.5 [10.7 to 41.2] | 53.3 [34.3 to 71.7] | 14.8 [4.2 to 33.7] | 5.6 [0.7 to 18.7] | 39.4 [22.9 to 57.9] | 23.3 [9.9 to 42.3] | 8.8 [1.9 to 23.7] | 21.2 [9.0 to 38.9] | 0 [0.0 to 10.3]
  M14: number analyzed (Participants) | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  M14 | 20 [8.4 to 36.9] | 25 [11.5 to 43.4] | 50 [29.9 to 70.1] | 30.8 [14.3 to 51.8] | 9.7 [2.0 to 25.8] | 38.7 [21.8 to 57.8] | 12 [2.5 to 31.2] | 3.3 [0.1 to 17.2] | 13.3 [3.8 to 30.7] | 0 [0.0 to 11.2]
  M14+28 days: number analyzed (Participants) | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  M14+28 days | 46.4 [27.5 to 66.1] | 83.9 [66.3 to 94.5] | 82.6 [61.2 to 95.0] | 44 [24.4 to 65.1] | 69 [49.2 to 84.7] | 75.9 [56.5 to 89.7] | 22.7 [7.8 to 45.4] | 38.5 [20.2 to 59.4] | 33.3 [16.5 to 54.0] | 10.3 [2.2 to 27.4]
  M20: number analyzed (Participants) | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  M20 | 27.6 [12.7 to 47.2] | 60 [40.6 to 77.3] | 50 [29.1 to 70.9] | 33.3 [15.6 to 55.3] | 38.7 [21.8 to 57.8] | 48.1 [28.7 to 68.1] | 20 [5.7 to 43.7] | 11.1 [2.4 to 29.2] | 25.9 [11.1 to 46.3] | 0 [0.0 to 13.7]
  M26: number analyzed (Participants) | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  M26 | 20.7 [8.0 to 39.7] | 41.4 [23.5 to 61.1] | 36.4 [17.2 to 59.3] | 28.6 [11.3 to 52.2] | 32 [14.9 to 53.5] | 36 [18.0 to 57.5] | 15 [3.2 to 37.9] | 8 [1.0 to 26.0] | 24 [9.4 to 45.1] | 0 [0.0 to 14.8]

44. Secondary Outcome: Percentage of Subjects With a ≥ 10-fold Increase of Anti-H1 Stalk Antibody Concentration, Measured by ELISA - Month 8 to 26.
Description: as for outcome 32
Time Frame: At Month 8, Month 14, Month 14 + 28 days, Month 20 and Month 26, compared to Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
Percentage of subjects
  M8 | 7.7 [1.6 to 20.9] | 0 [0.0 to 10.3] | 23.3 [9.9 to 42.3] | 7.4 [0.9 to 24.3] | 0 [0.0 to 9.7] | 9.1 [1.9 to 24.3] | 10 [2.1 to 26.5] | 0 [0.0 to 10.3] | 9.1 [1.9 to 24.3] | 0 [0.0 to 10.3]
  M14: number analyzed (Participants) | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  M14 | 5.7 [0.7 to 19.2] | 3.1 [0.1 to 16.2] | 30.8 [14.3 to 51.8] | 3.8 [0.1 to 19.6] | 3.2 [0.1 to 16.7] | 3.2 [0.1 to 16.7] | 4 [0.1 to 20.4] | 0 [0.0 to 11.6] | 10 [2.1 to 26.5] | 0 [0.0 to 11.2]
  M14+28 days: number analyzed (Participants) | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  M14+28 days | 17.9 [6.1 to 36.9] | 58.1 [39.1 to 75.5] | 52.2 [30.6 to 73.2] | 24 [9.4 to 45.1] | 37.9 [20.7 to 57.7] | 34.5 [17.9 to 54.3] | 4.5 [0.1 to 22.8] | 11.5 [2.4 to 30.2] | 18.5 [6.3 to 38.1] | 0 [0.0 to 11.9]
  M20: number analyzed (Participants) | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  M20 | 10.3 [2.2 to 27.4] | 26.7 [12.3 to 45.9] | 16.7 [4.7 to 37.4] | 8.3 [1.0 to 27.0] | 9.7 [2.0 to 25.8] | 11.1 [2.4 to 29.2] | 5 [0.1 to 24.9] | 3.7 [0.1 to 19.0] | 11.1 [2.4 to 29.2] | 0 [0.0 to 13.7]
  M26: number analyzed (Participants) | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  M26 | 3.4 [0.1 to 17.8] | 13.8 [3.9 to 31.7] | 4.5 [0.1 to 22.8] | 4.8 [0.1 to 23.8] | 4 [0.1 to 20.4] | 12 [2.5 to 31.2] | 10 [1.2 to 31.7] | 4 [0.1 to 20.4] | 12 [2.5 to 31.2] | 0 [0.0 to 14.8]

45. Secondary Outcome: MGI for Anti-H1 Stalk Antibody Measured by ELISA - Month 8 to 26
Description: MGI is defined as the geometric mean of the fold increase in serum HI concentration post-vaccination compared to Day 1
Time Frame: At Month 8, Month 14, Month 14 + 28 days, Month 20 and Month 26, compared to Day 1
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
Ratio
  M8 | 2.9 [2.2 to 3.7] | 2.3 [1.8 to 2.9] | 4.7 [3.5 to 6.3] | 2 [1.4 to 2.8] | 1.4 [1.2 to 1.8] | 3.3 [2.6 to 4.3] | 2.2 [1.5 to 3.1] | 1.3 [1.1 to 1.7] | 2.4 [1.7 to 3.3] | 1.3 [1.1 to 1.5]
  M14: number analyzed (Participants) | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  M14 | 2.5 [2.0 to 3.2] | 2.4 [1.8 to 3.2] | 4.7 [3.2 to 6.8] | 2.3 [1.7 to 3.2] | 1.6 [1.2 to 2.1] | 3.2 [2.5 to 4.2] | 2 [1.4 to 2.8] | 1.2 [1.0 to 1.5] | 2.1 [1.4 to 3.1] | 1.2 [1.0 to 1.4]
  M14+28 days: number analyzed (Participants) | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  M14+28 days | 5.3 [3.7 to 7.7] | 12.6 [8.7 to 18.2] | 9.5 [6.6 to 13.6] | 4.3 [3.0 to 6.4] | 7.3 [5.0 to 10.7] | 7.1 [5.3 to 9.5] | 2.7 [2.0 to 3.8] | 3.4 [2.3 to 5.0] | 4.1 [2.6 to 6.3] | 1.7 [1.3 to 2.2]
  M20: number analyzed (Participants) | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  M20 | 3 [2.3 to 3.8] | 4.9 [3.5 to 6.8] | 4.6 [3.3 to 6.3] | 2.6 [1.8 to 3.8] | 3.1 [2.3 to 4.1] | 4 [3.0 to 5.3] | 2.2 [1.5 to 3.2] | 1.8 [1.4 to 2.3] | 2.5 [1.7 to 3.6] | 1.3 [1.1 to 1.6]
  M26: number analyzed (Participants) | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  M26 | 2.7 [2.0 to 3.5] | 3.7 [2.7 to 5.2] | 3.7 [2.7 to 5.2] | 2.3 [1.5 to 3.6] | 2.6 [1.9 to 3.7] | 3.3 [2.4 to 4.4] | 2.1 [1.4 to 3.3] | 1.5 [1.1 to 2.1] | 2.2 [1.5 to 3.3] | 1.3 [1.1 to 1.6]

46. Secondary Outcome: Concentrations of Anti-H2 and Anti-H18 Antibodies Measured by ELISA
Description: Concentrations are presented as GMCs and measured by ELISA. ELISA cut-off = 22 EL.U/mL (H2) and 43 EL.U/mL (H18).
Time Frame: At Days 1, 29, 85, Month 8, Month 14, Month 14 + 28 days, Month 20 and Month 26
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 45 | 46 | 47 | 47 | 48 | 47 | 47 | 46 | 44 | 45
EL.U/mL
  Anti-H2, Day 1 | 5848.2 [4577.0 to 7472.5] | 5975.5 [4615.6 to 7736.1] | 6882.1 [5488.8 to 8629.2] | 5968.7 [4723.0 to 7542.9] | 6704 [5329.0 to 8433.8] | 5513.6 [4551.7 to 6678.7] | 6042.3 [4790.1 to 7622.0] | 5917.2 [4681.7 to 7478.9] | 6320.1 [4858.6 to 8221.2] | 5512.2 [4373.1 to 6948.0]
  Anti-H2, Day 29: number analyzed (Participants) | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
  Anti-H2, Day 29 | 111973.1 [90350.2 to 138770.8] | 28538 [22181.5 to 36716.0] | 115020.5 [93922.9 to 140857.1] | 59190.1 [46420.7 to 75472.2] | 30980 [25025.9 to 38350.8] | 64182.7 [50875.4 to 80970.8] | 30976.4 [20643.7 to 46481.0] | 12700 [10182.5 to 15839.8] | 33198.1 [25465.3 to 43279.1] | 10941.3 [8962.2 to 13357.5]
  Anti-H2, Day 85: number analyzed (Participants) | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
  Anti-H2, Day 85 | 42295.4 [34505.4 to 51844.2] | 18172.7 [13948.3 to 23676.6] | 60609.1 [47899.9 to 76690.5] | 26581.4 [19839.5 to 35614.4] | 16519.5 [13127.6 to 20787.9] | 39576.4 [31245.9 to 50128.0] | 23576.8 [15654.3 to 35508.7] | 9640.8 [7382.5 to 12590.1] | 29437.8 [22555.8 to 38419.7] | 8939.2 [7063.2 to 11313.4]
  Anti-H2, M8: number analyzed (Participants) | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
  Anti-H2, M8 | 29904.9 [24015.3 to 37238.9] | 12923.2 [9816.8 to 17012.6] | 38258.4 [29536.3 to 49556.3] | 18259.9 [13789.8 to 24179.0] | 12402.4 [9535.4 to 16131.4] | 24555.6 [19235.1 to 31347.7] | 19264.5 [13044.6 to 28450.1] | 8229 [6456.6 to 10488.1] | 22379.6 [17763.5 to 28195.2] | 9409 [7202.0 to 12292.4]
  Anti-H2, M14: number analyzed (Participants) | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  Anti-H2, M14 | 21754.4 [17375.9 to 27236.2] | 11417.4 [8969.1 to 14534.0] | 30670.3 [23748.7 to 39609.2] | 17100.4 [12454.3 to 23479.8] | 10899.7 [8122.1 to 14627.2] | 19573.6 [14935.3 to 25652.3] | 15050.2 [9969.1 to 22721.0] | 7717.7 [5839.8 to 10199.6] | 21978.5 [17171.0 to 28132.1] | 8582.5 [6443.9 to 11430.8]
  Anti-H2, M14+28 days: number analyzed (Participants) | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  Anti-H2, M14+28 days | 36459.1 [29419.5 to 45183.3] | 91778 [73053.9 to 115301.3] | 76909.5 [63594.4 to 93012.4] | 27256.3 [20573.9 to 36109.3] | 81616.2 [64374.2 to 103476.4] | 58542.1 [47219.6 to 72579.5] | 19172.9 [12543.2 to 29306.6] | 29940.3 [20765.3 to 43169.3] | 41953 [34398.2 to 51167.0] | 11753.1 [9023.9 to 15307.8]
  Anti-H2, M20: number analyzed (Participants) | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  Anti-H2, M20 | 24198.7 [19291.6 to 30353.9] | 34266 [26622.0 to 44104.8] | 36950 [29306.1 to 46587.6] | 19456.7 [14167.4 to 26720.7] | 32287.4 [25257.3 to 41274.2] | 28818 [22130.7 to 37525.9] | 14269 [9295.0 to 21905.0] | 15780.8 [11287.6 to 22062.7] | 25006.7 [19478.3 to 32104.2] | 7961.8 [5712.7 to 11096.2]
  Anti-H2, M26: number analyzed (Participants) | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  Anti-H2, M26 | 20136.5 [16257.6 to 24940.8] | 27000.7 [21059.5 to 34617.9] | 29403.8 [22530.7 to 38373.5] | 15358.6 [11070.7 to 21307.3] | 27477.2 [20295.7 to 37199.7] | 22917.6 [17205.8 to 30525.6] | 14906.4 [9433.3 to 23554.9] | 13186.7 [9162.6 to 18978.2] | 23570.6 [18496.4 to 30036.9] | 7708.3 [5593.3 to 10623.1]
  Anti-H18, Day 1: number analyzed (Participants) | 45 | 46 | 46 | 47 | 48 | 47 | 47 | 46 | 44 | 45
  Anti-H18, Day 1 | 4936.1 [3878.3 to 6282.3] | 4845.1 [3641.3 to 6446.9] | 5936.9 [4557.4 to 7734.1] | 5299.3 [4197.0 to 6691.1] | 5368.1 [4259.0 to 6766.0] | 4651.7 [3734.8 to 5793.7] | 4991.2 [4039.5 to 6167.0] | 5543.3 [4394.6 to 6992.4] | 5399.2 [4075.9 to 7152.3] | 5681.1 [4327.4 to 7458.4]
  Anti-H18, Day 29: number analyzed (Participants) | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
  Anti-H18, Day 29 | 26663.7 [21555.9 to 32981.8] | 19762.5 [15199.9 to 25694.6] | 30387.7 [25266.3 to 36547.2] | 19951 [16410.4 to 24255.6] | 21416.3 [17539.0 to 26150.8] | 19348 [16009.2 to 23383.0] | 13383.5 [9734.9 to 18399.5] | 10899.9 [8829.7 to 13455.5] | 14152.1 [11530.1 to 17370.3] | 11675.5 [9209.8 to 14801.4]
  Anti-H18, Day 85: number analyzed (Participants) | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
  Anti-H18, Day 85 | 13071 [10618.2 to 16090.3] | 13472.1 [10474.3 to 17327.9] | 27305.6 [22369.5 to 33330.8] | 10270.7 [8541.1 to 12350.5] | 12017.1 [9474.7 to 15241.8] | 17205.7 [14796.1 to 20007.7] | 10062.6 [7439.9 to 13610.1] | 8762.3 [6910.2 to 11110.9] | 15219.4 [12301.2 to 18829.9] | 9136.2 [6966.1 to 11982.3]
  Anti-H18, M8: number analyzed (Participants) | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
  Anti-H18, M8 | 11992.9 [9665.8 to 14880.2] | 10240.6 [7932.7 to 13220.0] | 18529.9 [15273.7 to 22480.4] | 10260.8 [8094.5 to 13006.8] | 9973.8 [7709.1 to 12903.9] | 12753.8 [10434.4 to 15588.8] | 9988.8 [7297.7 to 13672.3] | 8182.1 [6517.6 to 10271.7] | 12617.3 [10198.5 to 15609.8] | 9590.3 [7160.5 to 12844.6]
  Anti-H18, M14: number analyzed (Participants) | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  Anti-H18, M14 | 9039.6 [7212.3 to 11329.9] | 8610.3 [6938.0 to 10685.6] | 14078.6 [11455.9 to 17301.7] | 8820.4 [6959.4 to 11179.1] | 8370.2 [6213.2 to 11276.0] | 10216.5 [8035.8 to 12989.1] | 8526.2 [6047.8 to 12020.2] | 6955.8 [5553.1 to 8713.0] | 11876.7 [9622.1 to 14659.6] | 8178.4 [6007.8 to 11133.2]
  Anti-H18, M14+28 days: number analyzed (Participants) | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  Anti-H18, M14+28 days | 19763.3 [15225.3 to 25653.9] | 26567.6 [21331.9 to 33088.4] | 20291 [17142.5 to 24017.8] | 15768 [12672.2 to 19620.0] | 24020.6 [19157.0 to 30118.9] | 15872.3 [12888.2 to 19547.3] | 11742.6 [8553.4 to 16120.9] | 12543.5 [9593.4 to 16400.7] | 14564 [12163.0 to 17439.0] | 10758.1 [8190.4 to 14130.7]
  Anti-H18, M20: number analyzed (Participants) | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  Anti-H18, M20 | 12192 [9446.1 to 15736.1] | 14228.2 [11276.5 to 17952.5] | 13068.8 [10894.9 to 15676.5] | 10503.1 [8169.3 to 13503.6] | 12541.2 [9836.1 to 15990.2] | 10695.2 [8464.7 to 13513.5] | 9695.4 [6545.1 to 14362.2] | 8934.7 [6832.5 to 11683.6] | 12302.2 [9853.6 to 15359.2] | 7764.5 [5518.3 to 10925.1]
  Anti-H18, M26: number analyzed (Participants) | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  Anti-H18, M26 | 10832.8 [8488.3 to 13825.0] | 11823.4 [9575.2 to 14599.4] | 12186.4 [9948.2 to 14928.2] | 9767.9 [7407.6 to 12880.1] | 11445.8 [8371.9 to 15648.3] | 9308.8 [7285.1 to 11894.6] | 10283.6 [6627.6 to 15956.4] | 7937 [5903.9 to 10670.1] | 11617.9 [8948.6 to 15083.3] | 7646.4 [5326.5 to 10976.9]

47. Secondary Outcome: Number of Seropositive Subjects for Anti-H2 and Anti-H18 Antibodies Measured by ELISA
Description: Anti-H2 and anti-H18 immune response measured by ELISA. A seropositive subject is a subject whose concentration is greater than or equal to the cut-off value: ELISA cut-off = 22 EL.U/mL (H2) and 43 EL.U/mL (H18).
Time Frame: At Days 1, 29, 85, Month 8, Month 14, Month 14 + 28 days, Month 20 and Month 26
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 45 | 46 | 47 | 47 | 48 | 47 | 47 | 46 | 44 | 45
Participants
  Anti-H2, Day 1 | 45 | 46 | 47 | 47 | 48 | 47 | 47 | 46 | 44 | 45
  Anti-H2, Day 29: number analyzed (Participants) | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
  Anti-H2, Day 29 | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
  Anti-H2, Day 85: number analyzed (Participants) | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
  Anti-H2, Day 85 | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
  Anti-H2, M8: number analyzed (Participants) | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
  Anti-H2, M8 | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
  Anti-H2, M14: number analyzed (Participants) | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  Anti-H2, M14 | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  Anti-H2, M14+28 days: number analyzed (Participants) | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  Anti-H2, M14+28 days | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  Anti-H2, M20: number analyzed (Participants) | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  Anti-H2, M20 | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  Anti-H2, M26: number analyzed (Participants) | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  Anti-H2, M26 | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  Anti-H18, Day 1: number analyzed (Participants) | 45 | 46 | 46 | 47 | 48 | 47 | 47 | 46 | 44 | 45
  Anti-H18, Day 1 | 45 | 46 | 46 | 47 | 48 | 47 | 47 | 46 | 44 | 45
  Anti-H18, Day 29: number analyzed (Participants) | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
  Anti-H18, Day 29 | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
  Anti-H18, Day 85: number analyzed (Participants) | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
  Anti-H18, Day 85 | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
  Anti-H18, M8: number analyzed (Participants) | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
  Anti-H18, M8 | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
  Anti-H18, M14: number analyzed (Participants) | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  Anti-H18, M14 | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  Anti-H18, M14+28 days: number analyzed (Participants) | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  Anti-H18, M14+28 days | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  Anti-H18, M20: number analyzed (Participants) | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  Anti-H18, M20 | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  Anti-H18, M26: number analyzed (Participants) | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  Anti-H18, M26 | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23

48. Secondary Outcome: Percentage of Subjects With a ≥ 4-fold Increase of Anti-H2 and Anti-H18 Antibody Concentration Measured by ELISA
Description: Percentage of subjects with a ≥ 4-fold increase of anti-H2 and anti-H18 antibody concentration, from Day 1, is calculated with exact 95% CI by ELISA .
Time Frame: At Day 29, at Day 85, Month 8, Month 14, Month 14 + 28 days, Month 20 and Month 26, compared to Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
Percentage of subjects
  Anti-H2, Day 29 | 95.3 [84.2 to 99.4] | 62.5 [45.8 to 77.3] | 92.7 [80.1 to 98.5] | 82.5 [67.2 to 92.7] | 57.1 [41.0 to 72.3] | 90.5 [77.4 to 97.3] | 62.2 [44.8 to 77.5] | 26.8 [14.2 to 42.9] | 48.7 [32.4 to 65.2] | 12.5 [4.2 to 26.8]
  Anti-H2, Day 85: number analyzed (Participants) | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
  Anti-H2, Day 85 | 66.7 [49.8 to 80.9] | 36.1 [20.8 to 53.8] | 79.4 [62.1 to 91.3] | 45.7 [28.8 to 63.4] | 17.9 [7.5 to 33.5] | 77.1 [59.9 to 89.6] | 35.3 [19.7 to 53.5] | 2.9 [0.1 to 15.3] | 42.9 [26.3 to 60.6] | 5.3 [0.6 to 17.7]
  Anti-H2, M8: number analyzed (Participants) | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
  Anti-H2, M8 | 51.3 [34.8 to 67.6] | 23.5 [10.7 to 41.2] | 73.3 [54.1 to 87.7] | 29.6 [13.8 to 50.2] | 8.3 [1.8 to 22.5] | 69.7 [51.3 to 84.4] | 26.7 [12.3 to 45.9] | 5.9 [0.7 to 19.7] | 33.3 [18.0 to 51.8] | 0 [0.0 to 10.3]
  Anti-H2, M14: number analyzed (Participants) | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  Anti-H2, M14 | 34.3 [19.1 to 52.2] | 15.6 [5.3 to 32.8] | 61.5 [40.6 to 79.8] | 30.8 [14.3 to 51.8] | 6.5 [0.8 to 21.4] | 58.1 [39.1 to 75.5] | 16 [4.5 to 36.1] | 3.3 [0.1 to 17.2] | 23.3 [9.9 to 42.3] | 0 [0.0 to 11.2]
  Anti-H2, M14+28 days: number analyzed (Participants) | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  Anti-H2, M14+28 days | 57.1 [37.2 to 75.5] | 100 [88.8 to 100.0] | 100 [85.2 to 100.0] | 52 [31.3 to 72.2] | 82.8 [64.2 to 94.2] | 96.6 [82.2 to 99.9] | 36.4 [17.2 to 59.3] | 50 [29.9 to 70.1] | 63 [42.4 to 80.6] | 6.9 [0.8 to 22.8]
  Anti-H2, M20: number analyzed (Participants) | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  Anti-H2, M20 | 41.4 [23.5 to 61.1] | 70 [50.6 to 85.3] | 75 [53.3 to 90.2] | 41.7 [22.1 to 63.4] | 54.8 [36.0 to 72.7] | 74.1 [53.7 to 88.9] | 20 [5.7 to 43.7] | 18.5 [6.3 to 38.1] | 37 [19.4 to 57.6] | 4 [0.1 to 20.4]
  Anti-H2, M26: number analyzed (Participants) | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  Anti-H2, M26 | 41.4 [23.5 to 61.1] | 62.1 [42.3 to 79.3] | 54.5 [32.2 to 75.6] | 38.1 [18.1 to 61.6] | 48 [27.8 to 68.7] | 56 [34.9 to 75.6] | 20 [5.7 to 43.7] | 16 [4.5 to 36.1] | 32 [14.9 to 53.5] | 4.3 [0.1 to 21.9]
  Anti-H18, Day 29: number analyzed (Participants) | 43 | 40 | 40 | 40 | 42 | 42 | 37 | 41 | 39 | 40
  Anti-H18, Day 29 | 55.8 [39.9 to 70.9] | 52.5 [36.1 to 68.5] | 50 [33.8 to 66.2] | 40 [24.9 to 56.7] | 45.2 [29.8 to 61.3] | 52.4 [36.4 to 68.0] | 21.6 [9.8 to 38.2] | 19.5 [8.8 to 34.9] | 20.5 [9.3 to 36.5] | 15 [5.7 to 29.8]
  Anti-H18, Day 85: number analyzed (Participants) | 39 | 36 | 33 | 35 | 39 | 35 | 34 | 34 | 35 | 38
  Anti-H18, Day 85 | 17.9 [7.5 to 33.5] | 33.3 [18.6 to 51.0] | 48.5 [30.8 to 66.5] | 14.3 [4.8 to 30.3] | 20.5 [9.3 to 36.5] | 48.6 [31.4 to 66.0] | 14.7 [5.0 to 31.1] | 5.9 [0.7 to 19.7] | 25.7 [12.5 to 43.3] | 5.3 [0.6 to 17.7]
  Anti-H18, M8: number analyzed (Participants) | 39 | 34 | 29 | 27 | 36 | 33 | 30 | 34 | 33 | 34
  Anti-H18, M8 | 12.8 [4.3 to 27.4] | 20.6 [8.7 to 37.9] | 44.8 [26.4 to 64.3] | 11.1 [2.4 to 29.2] | 11.1 [3.1 to 26.1] | 39.4 [22.9 to 57.9] | 16.7 [5.6 to 34.7] | 11.8 [3.3 to 27.5] | 24.2 [11.1 to 42.3] | 0 [0.0 to 10.3]
  Anti-H18, M14: number analyzed (Participants) | 35 | 32 | 25 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  Anti-H18, M14 | 8.6 [1.8 to 23.1] | 21.9 [9.3 to 40.0] | 36 [18.0 to 57.5] | 11.5 [2.4 to 30.2] | 6.5 [0.8 to 21.4] | 29 [14.2 to 48.0] | 8 [1.0 to 26.0] | 3.3 [0.1 to 17.2] | 13.3 [3.8 to 30.7] | 0 [0.0 to 11.2]
  Anti-H18, M14+28 days: number analyzed (Participants) | 28 | 31 | 22 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  Anti-H18, M14+28 days | 35.7 [18.6 to 55.9] | 71 [52.0 to 85.8] | 54.5 [32.2 to 75.6] | 36 [18.0 to 57.5] | 55.2 [35.7 to 73.6] | 55.2 [35.7 to 73.6] | 18.2 [5.2 to 40.3] | 15.4 [4.4 to 34.9] | 25.9 [11.1 to 46.3] | 6.9 [0.8 to 22.8]
  Anti-H18, M20: number analyzed (Participants) | 29 | 30 | 23 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  Anti-H18, M20 | 20.7 [8.0 to 39.7] | 40 [22.7 to 59.4] | 30.4 [13.2 to 52.9] | 20.8 [7.1 to 42.2] | 19.4 [7.5 to 37.5] | 29.6 [13.8 to 50.2] | 5 [0.1 to 24.9] | 7.4 [0.9 to 24.3] | 11.1 [2.4 to 29.2] | 4 [0.1 to 20.4]
  Anti-H18, M26: number analyzed (Participants) | 29 | 29 | 21 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  Anti-H18, M26 | 24.1 [10.3 to 43.5] | 31 [15.3 to 50.8] | 28.6 [11.3 to 52.2] | 23.8 [8.2 to 47.2] | 20 [6.8 to 40.7] | 12 [2.5 to 31.2] | 10 [1.2 to 31.7] | 8 [1.0 to 26.0] | 12 [2.5 to 31.2] | 0 [0.0 to 14.8]

49. Secondary Outcome: Percentage of Subjects With a ≥ 10-fold Increase of Anti-H2 and Anti-H18 Antibody Concentration Measured by ELISA
Description: Percentage of subjects with a ≥ 10-fold increase of anti-H2 and anti-H18 antibody concentration, from Day 1, is calculated with exact 95% CI by ELISA .
Time Frame: At Day 29, at Day 85, Month 8, Month 14, Month 14 + 28 days, Month 20 and Month 26, compared to Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
Percentage of subjects
  Anti-H2, Day 29 | 67.4 [51.5 to 80.9] | 15 [5.7 to 29.8] | 68.3 [51.9 to 81.9] | 42.5 [27.0 to 59.1] | 16.7 [7.0 to 31.4] | 61.9 [45.6 to 76.4] | 18.9 [8.0 to 35.2] | 2.4 [0.1 to 12.9] | 20.5 [9.3 to 36.5] | 2.5 [0.1 to 13.2]
  Anti-H2, Day 85: number analyzed (Participants) | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
  Anti-H2, Day 85 | 25.6 [13.0 to 42.1] | 5.6 [0.7 to 18.7] | 55.9 [37.9 to 72.8] | 22.9 [10.4 to 40.1] | 2.6 [0.1 to 13.5] | 48.6 [31.4 to 66.0] | 20.6 [8.7 to 37.9] | 2.9 [0.1 to 15.3] | 17.1 [6.6 to 33.6] | 5.3 [0.6 to 17.7]
  Anti-H2, M8: number analyzed (Participants) | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
  Anti-H2, M8 | 15.4 [5.9 to 30.5] | 0 [0.0 to 10.3] | 26.7 [12.3 to 45.9] | 11.1 [2.4 to 29.2] | 0 [0.0 to 9.7] | 12.1 [3.4 to 28.2] | 16.7 [5.6 to 34.7] | 0 [0.0 to 10.3] | 15.2 [5.1 to 31.9] | 0 [0.0 to 10.3]
  Anti-H2, M14: number analyzed (Participants) | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  Anti-H2, M14 | 14.3 [4.8 to 30.3] | 0 [0.0 to 10.9] | 23.1 [9.0 to 43.6] | 11.5 [2.4 to 30.2] | 0 [0.0 to 11.2] | 6.5 [0.8 to 21.4] | 8 [1.0 to 26.0] | 0 [0.0 to 11.6] | 10 [2.1 to 26.5] | 0 [0.0 to 11.2]
  Anti-H2, M14+28 days: number analyzed (Participants) | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  Anti-H2, M14+28 days | 25 [10.7 to 44.9] | 71 [52.0 to 85.8] | 65.2 [42.7 to 83.6] | 24 [9.4 to 45.1] | 48.3 [29.4 to 67.5] | 65.5 [45.7 to 82.1] | 9.1 [1.1 to 29.2] | 15.4 [4.4 to 34.9] | 22.2 [8.6 to 42.3] | 3.4 [0.1 to 17.8]
  Anti-H2, M20: number analyzed (Participants) | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  Anti-H2, M20 | 13.8 [3.9 to 31.7] | 23.3 [9.9 to 42.3] | 25 [9.8 to 46.7] | 20.8 [7.1 to 42.2] | 25.8 [11.9 to 44.6] | 22.2 [8.6 to 42.3] | 5 [0.1 to 24.9] | 7.4 [0.9 to 24.3] | 11.1 [2.4 to 29.2] | 0 [0.0 to 13.7]
  Anti-H2, M26: number analyzed (Participants) | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  Anti-H2, M26 | 13.8 [3.9 to 31.7] | 13.8 [3.9 to 31.7] | 18.2 [5.2 to 40.3] | 9.5 [1.2 to 30.4] | 24 [9.4 to 45.1] | 12 [2.5 to 31.2] | 10 [1.2 to 31.7] | 8 [1.0 to 26.0] | 12 [2.5 to 31.2] | 0 [0.0 to 14.8]
  Anti-H18, Day 29: number analyzed (Participants) | 43 | 40 | 40 | 40 | 42 | 42 | 37 | 41 | 39 | 40
  Anti-H18, Day 29 | 23.3 [11.8 to 38.6] | 15 [5.7 to 29.8] | 25 [12.7 to 41.2] | 12.5 [4.2 to 26.8] | 16.7 [7.0 to 31.4] | 16.7 [7.0 to 31.4] | 8.1 [1.7 to 21.9] | 2.4 [0.1 to 12.9] | 7.7 [1.6 to 20.9] | 2.5 [0.1 to 13.2]
  Anti-H18, Day 85: number analyzed (Participants) | 39 | 36 | 33 | 35 | 39 | 35 | 34 | 34 | 35 | 38
  Anti-H18, Day 85 | 7.7 [1.6 to 20.9] | 2.8 [0.1 to 14.5] | 24.2 [11.1 to 42.3] | 5.7 [0.7 to 19.2] | 2.6 [0.1 to 13.5] | 5.7 [0.7 to 19.2] | 2.9 [0.1 to 15.3] | 2.9 [0.1 to 15.3] | 11.4 [3.2 to 26.7] | 5.3 [0.6 to 17.7]
  Anti-H18, M8: number analyzed (Participants) | 39 | 34 | 29 | 27 | 36 | 33 | 30 | 34 | 33 | 34
  Anti-H18, M8 | 2.6 [0.1 to 13.5] | 0 [0.0 to 10.3] | 6.9 [0.8 to 22.8] | 3.7 [0.1 to 19.0] | 0 [0.0 to 9.7] | 3 [0.1 to 15.8] | 6.7 [0.8 to 22.1] | 2.9 [0.1 to 15.3] | 9.1 [1.9 to 24.3] | 0 [0.0 to 10.3]
  Anti-H18, M14: number analyzed (Participants) | 35 | 32 | 25 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  Anti-H18, M14 | 0 [0.0 to 10.0] | 0 [0.0 to 10.9] | 12 [2.5 to 31.2] | 3.8 [0.1 to 19.6] | 0 [0.0 to 11.2] | 0 [0.0 to 11.2] | 4 [0.1 to 20.4] | 0 [0.0 to 11.6] | 10 [2.1 to 26.5] | 0 [0.0 to 11.2]
  Anti-H18, M14+28 days: number analyzed (Participants) | 28 | 31 | 22 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  Anti-H18, M14+28 days | 17.9 [6.1 to 36.9] | 25.8 [11.9 to 44.6] | 18.2 [5.2 to 40.3] | 12 [2.5 to 31.2] | 17.2 [5.8 to 35.8] | 3.4 [0.1 to 17.8] | 4.5 [0.1 to 22.8] | 7.7 [0.9 to 25.1] | 11.1 [2.4 to 29.2] | 0 [0.0 to 11.9]
  Anti-H18, M20: number analyzed (Participants) | 29 | 30 | 23 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  Anti-H18, M20 | 6.9 [0.8 to 22.8] | 13.3 [3.8 to 30.7] | 4.3 [0.1 to 21.9] | 4.2 [0.1 to 21.1] | 6.5 [0.8 to 21.4] | 0 [0.0 to 12.8] | 5 [0.1 to 24.9] | 3.7 [0.1 to 19.0] | 11.1 [2.4 to 29.2] | 0 [0.0 to 13.7]
  Anti-H18, M26: number analyzed (Participants) | 29 | 29 | 21 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  Anti-H18, M26 | 6.9 [0.8 to 22.8] | 10.3 [2.2 to 27.4] | 4.8 [0.1 to 23.8] | 4.8 [0.1 to 23.8] | 8 [1.0 to 26.0] | 0 [0.0 to 13.7] | 10 [1.2 to 31.7] | 0 [0.0 to 13.7] | 8 [1.0 to 26.0] | 0 [0.0 to 14.8]

50. Secondary Outcome: MGI for Anti-H2 and Anti-H18 Antibodies Concentrations Measured by ELISA
Description: MGI is defined as the geometric mean of the fold increase in serum HI concentration post-vaccination compared to Day 1.
Time Frame: At Day 29, at Day 85, Month 8, Month 14, Month 14 + 28 days, Month 20 and Month 26, compared to Day 1
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 41 | 40 | 42 | 42 | 37 | 41 | 39 | 40
Ratio
  Anti-H2, Day 29 | 18.4 [13.6 to 24.9] | 5.3 [4.0 to 7.0] | 17.3 [12.9 to 23.1] | 9.9 [7.0 to 14.0] | 4.7 [3.7 to 6.0] | 12.3 [9.2 to 16.3] | 5.6 [3.8 to 8.1] | 2.3 [1.8 to 2.9] | 5 [3.5 to 7.0] | 1.9 [1.6 to 2.3]
  Anti-H2, Day 85: number analyzed (Participants) | 39 | 36 | 34 | 35 | 39 | 35 | 34 | 34 | 35 | 38
  Anti-H2, Day 85 | 7 [5.2 to 9.2] | 3.2 [2.5 to 4.2] | 9.5 [7.2 to 12.5] | 4.4 [3.0 to 6.5] | 2.4 [2.0 to 2.9] | 8.2 [6.3 to 10.7] | 4.1 [2.8 to 5.8] | 1.7 [1.4 to 2.0] | 4.2 [2.9 to 6.1] | 1.6 [1.3 to 1.9]
  Anti-H2, M8: number analyzed (Participants) | 39 | 34 | 30 | 27 | 36 | 33 | 30 | 34 | 33 | 34
  Anti-H2, M8 | 4.8 [3.7 to 6.2] | 2.4 [1.9 to 2.9] | 6.2 [4.6 to 8.4] | 3.1 [2.1 to 4.4] | 1.8 [1.5 to 2.1] | 5.2 [4.0 to 6.6] | 3.3 [2.2 to 4.9] | 1.5 [1.3 to 1.8] | 3.3 [2.3 to 4.7] | 1.5 [1.3 to 1.7]
  Anti-H2, M14: number analyzed (Participants) | 35 | 32 | 26 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  Anti-H2, M14 | 3.6 [2.8 to 4.7] | 2.2 [1.8 to 2.6] | 5.6 [3.9 to 8.1] | 3.1 [2.1 to 4.5] | 1.6 [1.4 to 2.0] | 4.1 [3.3 to 5.3] | 2.5 [1.8 to 3.6] | 1.4 [1.2 to 1.7] | 2.8 [2.0 to 4.0] | 1.4 [1.2 to 1.6]
  Anti-H2, M14+28 days: number analyzed (Participants) | 28 | 31 | 23 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  Anti-H2, M14+28 days | 6.1 [4.3 to 8.7] | 17.2 [12.5 to 23.8] | 14.7 [10.4 to 20.8] | 5.1 [3.4 to 7.7] | 12.1 [8.0 to 18.3] | 12.6 [9.7 to 16.2] | 3.3 [2.3 to 4.8] | 5.6 [3.7 to 8.4] | 6.1 [4.2 to 8.9] | 1.9 [1.5 to 2.3]
  Anti-H2, M20: number analyzed (Participants) | 29 | 30 | 24 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  Anti-H2, M20 | 3.9 [3.0 to 5.1] | 6.4 [4.8 to 8.7] | 6.5 [4.6 to 9.0] | 3.6 [2.4 to 5.3] | 4.8 [3.4 to 6.9] | 6.2 [4.8 to 8.0] | 2.5 [1.7 to 3.6] | 2.7 [1.9 to 3.9] | 3.7 [2.6 to 5.2] | 1.3 [1.1 to 1.6]
  Anti-H2, M26: number analyzed (Participants) | 29 | 29 | 22 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  Anti-H2, M26 | 3.5 [2.7 to 4.6] | 5 [3.7 to 6.7] | 5 [3.5 to 7.1] | 3 [2.0 to 4.7] | 4.2 [2.8 to 6.1] | 4.9 [3.7 to 6.5] | 2.6 [1.7 to 3.9] | 2.3 [1.6 to 3.4] | 3.2 [2.2 to 4.6] | 1.4 [1.2 to 1.6]
  Anti-H18, Day 29: number analyzed (Participants) | 43 | 40 | 40 | 40 | 42 | 42 | 37 | 41 | 39 | 40
  Anti-H18, Day 29 | 5.2 [3.9 to 6.9] | 4.6 [3.5 to 6.0] | 5.3 [3.8 to 7.3] | 3.7 [2.8 to 4.9] | 4.1 [3.2 to 5.3] | 4.3 [3.3 to 5.6] | 2.7 [2.0 to 3.7] | 2.1 [1.7 to 2.7] | 2.5 [1.9 to 3.3] | 2 [1.7 to 2.4]
  Anti-H18, Day 85: number analyzed (Participants) | 39 | 36 | 33 | 35 | 39 | 35 | 34 | 34 | 35 | 38
  Anti-H18, Day 85 | 2.6 [2.1 to 3.3] | 2.9 [2.2 to 3.7] | 4.9 [3.7 to 6.5] | 2 [1.5 to 2.7] | 2.2 [1.8 to 2.7] | 4.3 [3.4 to 5.3] | 2 [1.5 to 2.7] | 1.6 [1.4 to 2.0] | 2.6 [1.9 to 3.6] | 1.6 [1.3 to 1.9]
  Anti-H18, M8: number analyzed (Participants) | 39 | 34 | 29 | 27 | 36 | 33 | 30 | 34 | 33 | 34
  Anti-H18, M8 | 2.4 [1.9 to 2.9] | 2.4 [1.9 to 3.0] | 3.5 [2.6 to 4.6] | 1.8 [1.4 to 2.4] | 1.8 [1.5 to 2.2] | 3.2 [2.6 to 3.9] | 2 [1.5 to 2.7] | 1.6 [1.3 to 2.0] | 2.3 [1.7 to 3.2] | 1.5 [1.3 to 1.7]
  Anti-H18, M14: number analyzed (Participants) | 35 | 32 | 25 | 26 | 31 | 31 | 25 | 30 | 30 | 31
  Anti-H18, M14 | 1.9 [1.5 to 2.2] | 2.1 [1.7 to 2.6] | 3.1 [2.3 to 4.4] | 1.8 [1.3 to 2.4] | 1.6 [1.3 to 2.0] | 2.6 [2.1 to 3.3] | 1.7 [1.2 to 2.3] | 1.3 [1.1 to 1.5] | 1.9 [1.4 to 2.5] | 1.3 [1.1 to 1.5]
  Anti-H18, M14+28 days: number analyzed (Participants) | 28 | 31 | 22 | 25 | 29 | 29 | 22 | 26 | 27 | 29
  Anti-H18, M14+28 days | 4.1 [2.9 to 5.7] | 6.4 [4.6 to 9.0] | 4.6 [3.1 to 6.6] | 3.3 [2.3 to 4.7] | 4.4 [3.3 to 5.9] | 4.3 [3.4 to 5.3] | 2.4 [1.8 to 3.3] | 2.4 [1.8 to 3.2] | 2.6 [1.8 to 3.6] | 1.7 [1.3 to 2.1]
  Anti-H18, M20: number analyzed (Participants) | 29 | 30 | 23 | 24 | 31 | 27 | 20 | 27 | 27 | 25
  Anti-H18, M20 | 2.5 [1.9 to 3.1] | 3.5 [2.6 to 4.8] | 2.7 [2.0 to 3.8] | 2.2 [1.6 to 3.1] | 2.4 [1.9 to 3.1] | 2.8 [2.3 to 3.5] | 2 [1.4 to 2.8] | 1.6 [1.3 to 2.0] | 2.1 [1.6 to 2.9] | 1.3 [1.1 to 1.6]
  Anti-H18, M26: number analyzed (Participants) | 29 | 29 | 21 | 21 | 25 | 25 | 20 | 25 | 25 | 23
  Anti-H18, M26 | 2.4 [1.8 to 3.0] | 2.9 [2.1 to 3.9] | 2.4 [1.7 to 3.4] | 2.1 [1.5 to 3.1] | 2.2 [1.6 to 3.0] | 2.5 [2.0 to 3.1] | 2.1 [1.4 to 3.2] | 1.4 [1.1 to 1.8] | 1.9 [1.3 to 2.8] | 1.4 [1.2 to 1.6]

51. Secondary Outcome: Titers for Anti-H1N1 Swine Influenza and Anti-IIV4-H1N1 Anti-bodies Measured by MN Assay
Description: Titers are presented as GMTs and measured by MN assay. MN cut-off = 20 1/DIL
Time Frame: At Days 1, 29 and 85
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 45 | 46 | 46 | 46 | 47 | 47 | 47 | 46 | 44 | 45
Titer
  Day 1 | 58.8 [45.6 to 75.7] | 61 [47.8 to 77.8] | 62.9 [50.8 to 77.8] | 51.7 [39.5 to 67.6] | 53.7 [42.6 to 67.7] | 56.2 [44.5 to 70.8] | 56.2 [45.6 to 69.1] | 70.9 [57.3 to 87.8] | 56.6 [45.2 to 70.8] | 60.6 [48.9 to 75.2]
  Day 29: number analyzed (Participants) | 43 | 40 | 40 | 40 | 41 | 42 | 37 | 41 | 39 | 40
  Day 29 | 84 [68.8 to 102.5] | 93.5 [76.7 to 113.9] | 87.2 [77.0 to 98.8] | 84.3 [74.2 to 95.7] | 93.1 [82.2 to 105.5] | 80 [67.8 to 94.4] | 71.5 [59.4 to 86.0] | 78.7 [64.9 to 95.4] | 69.4 [54.1 to 88.9] | 103.7 [88.0 to 122.3]
  Day 85: number analyzed (Participants) | 39 | 36 | 34 | 35 | 38 | 35 | 34 | 34 | 35 | 38
  Day 85 | 65.8 [49.6 to 87.2] | 89.8 [73.7 to 109.5] | 96.1 [83.8 to 110.2] | 56 [45.3 to 69.2] | 81.5 [68.1 to 97.5] | 86.6 [73.7 to 101.7] | 63.9 [51.7 to 79.1] | 68 [52.8 to 87.5] | 84.9 [72.6 to 99.3] | 99.6 [78.5 to 126.3]

52. Secondary Outcome: Number of Seropositive Subjects for Anti-H1N1 Swine Influenza and Anti-IIV4-H1N1 Antibodies Measured by MN Assay
Description: Anti-H1N1 swine influenza and anti-IIV4-H1N1 immune response measured by MN assay. A seropositive subject is a subject whose titer is greater than or equal to the cut-off value: cut-off = 20 1/DIL.
Time Frame: At Days 1, 29 and 85
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 45 | 46 | 46 | 46 | 47 | 47 | 47 | 46 | 44 | 45
Participants
  Day 1 | 40 | 41 | 43 | 38 | 42 | 42 | 44 | 43 | 42 | 43
  Day 29: number analyzed (Participants) | 43 | 40 | 40 | 40 | 41 | 42 | 37 | 41 | 39 | 40
  Day 29 | 42 | 39 | 40 | 40 | 41 | 42 | 37 | 40 | 36 | 40
  Day 85: number analyzed (Participants) | 39 | 36 | 34 | 35 | 38 | 35 | 34 | 34 | 35 | 38
  Day 85 | 36 | 35 | 34 | 34 | 38 | 35 | 34 | 32 | 35 | 37

53. Secondary Outcome: Percentage of Subjects With a ≥ 4-fold Increase of Anti-H1N1 Swine Influenza and Anti-IIV4-H1N1 Antibody Titers Measured by MN Assay
Description: Percentage of subjects with a ≥ 4-fold increase of anti-H1N1 swine influenza and anti-IIV4-H1N1 antibody titers, from Day 1, is calculated with exact 95% CI by MN assay.
Time Frame: At Day 29 and Day 85, compared to Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 39 | 39 | 41 | 42 | 37 | 41 | 39 | 40
Percentage of subjects
  Day 29 | 9.3 [2.6 to 22.1] | 22.5 [10.8 to 38.5] | 7.7 [1.6 to 20.9] | 23.1 [11.1 to 39.3] | 24.4 [12.4 to 40.3] | 9.5 [2.7 to 22.6] | 10.8 [3.0 to 25.4] | 2.4 [0.1 to 12.9] | 7.7 [1.6 to 20.9] | 15 [5.7 to 29.8]
  Day 85: number analyzed (Participants) | 39 | 36 | 33 | 34 | 38 | 35 | 34 | 34 | 35 | 38
  Day 85 | 5.1 [0.6 to 17.3] | 16.7 [6.4 to 32.8] | 18.2 [7.0 to 35.5] | 5.9 [0.7 to 19.7] | 21.1 [9.6 to 37.3] | 14.3 [4.8 to 30.3] | 5.9 [0.7 to 19.7] | 0 [0.0 to 10.3] | 8.6 [1.8 to 23.1] | 15.8 [6.0 to 31.3]

54. Secondary Outcome: Percentage of Subjects With a ≥ 10-fold Increase of Anti-H1N1 Swine Influenza and Anti-IIV4-H1N1 Antibody Titers Measured by MN Assay
Description: Percentage of subjects with a ≥ 10-fold increase of anti-H1N1 swine influenza and anti-IIV4-H1N1 antibody titers, from Day 1, is calculated with exact 95% CI by MN assay.
Time Frame: At Day 29 and Day 85, compared to Day 1
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 39 | 39 | 41 | 42 | 37 | 41 | 39 | 40
Percentage of subjects
  Day 29 | 2.3 [0.1 to 12.3] | 2.5 [0.1 to 13.2] | 0 [0.0 to 9.0] | 0 [0.0 to 9.0] | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 9.5] | 0 [0.0 to 8.6] | 0 [0.0 to 9.0] | 0 [0.0 to 8.8]
  Day 85: number analyzed (Participants) | 39 | 36 | 33 | 34 | 38 | 35 | 34 | 34 | 35 | 38
  Day 85 | 0 [0.0 to 9.0] | 2.8 [0.1 to 14.5] | 3 [0.1 to 15.8] | 0 [0.0 to 10.3] | 0 [0.0 to 9.3] | 2.9 [0.1 to 14.9] | 0 [0.0 to 10.3] | 0 [0.0 to 10.3] | 0 [0.0 to 10.0] | 0 [0.0 to 9.3]

55. Secondary Outcome: MGI for Anti-H1N1 Swine Influenza and Anti-IIV4-H1N1 Antibodies Titers Measured by MN Assay
Description: MGI is defined as the geometric mean of the fold increase in serum HI titer post-vaccination compared to Day 1.
Time Frame: At Day 29 and at Day 85, compared to Day 1
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
Number analyzed (Participants) | 43 | 40 | 39 | 39 | 41 | 42 | 37 | 41 | 39 | 40
Ratio
  Day 29 | 1.4 [1.1 to 1.7] | 1.7 [1.3 to 2.1] | 1.4 [1.2 to 1.6] | 1.7 [1.3 to 2.2] | 1.7 [1.4 to 2.2] | 1.4 [1.2 to 1.7] | 1.3 [1.0 to 1.5] | 1.1 [0.9 to 1.3] | 1.2 [1.0 to 1.5] | 1.7 [1.4 to 2.0]
  Day 85: number analyzed (Participants) | 39 | 36 | 33 | 34 | 38 | 35 | 34 | 34 | 35 | 38
  Day 85 | 1.1 [0.9 to 1.3] | 1.5 [1.1 to 2.0] | 1.6 [1.2 to 2.1] | 1 [0.9 to 1.3] | 1.5 [1.2 to 1.9] | 1.5 [1.2 to 1.9] | 1.1 [0.9 to 1.3] | 0.9 [0.8 to 1.1] | 1.3 [1.1 to 1.6] | 1.5 [1.3 to 1.9]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected during the 7-day follow-up period after each vaccination. Unsolicited AEs were collected during the 28-day follow-up period after any vaccination. SAEs were collected during the entire study period (from Day 1 up to Month 26).
Arm/Group | D-SUIV Adjuvanted Group 1 | D-SUIV Adjuvanted Group 2 | D-SUIV Adjuvanted Group 3 | D-SUIV Adjuvanted Group 4 | D-SUIV Adjuvanted Group 5 | D-SUIV Adjuvanted Group 6 | D-SUIV Unadjuvanted Group 1 | D-SUIV Unadjuvanted Group 2 | D-SUIV Unadjuvanted Group 3 | IIV4 Group
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/46 | 0/47 | 0/47 | 0/48 | 1/47 | 0/47 | 0/48 | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 2/45 | 1/46 | 1/47 | 2/47 | 2/48 | 2/47 | 0/47 | 2/48 | 2/46 | 3/47
Other Adverse Events (participants affected / at risk) | 40/45 | 43/46 | 44/47 | 44/47 | 45/48 | 44/47 | 34/47 | 38/48 | 42/46 | 44/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-SUIV Adjuvanted Group 1 (N=45) | D-SUIV Adjuvanted Group 2 (N=46) | D-SUIV Adjuvanted Group 3 (N=47) | D-SUIV Adjuvanted Group 4 (N=47) | D-SUIV Adjuvanted Group 5 (N=48) | D-SUIV Adjuvanted Group 6 (N=47) | D-SUIV Unadjuvanted Group 1 (N=47) | D-SUIV Unadjuvanted Group 2 (N=48) | D-SUIV Unadjuvanted Group 3 (N=46) | IIV4 Group (N=47)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-SUIV Adjuvanted Group 1 (N=45) | D-SUIV Adjuvanted Group 2 (N=46) | D-SUIV Adjuvanted Group 3 (N=47) | D-SUIV Adjuvanted Group 4 (N=47) | D-SUIV Adjuvanted Group 5 (N=48) | D-SUIV Adjuvanted Group 6 (N=47) | D-SUIV Unadjuvanted Group 1 (N=47) | D-SUIV Unadjuvanted Group 2 (N=48) | D-SUIV Unadjuvanted Group 3 (N=46) | IIV4 Group (N=47)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 10 (12) | 15 (19) | 14 (22) | 11 (14) | 12 (17) | 15 (19) | 8 (8) | 10 (14) | 12 (16) | 9 (10)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 9 (13) | 16 (20) | 15 (20) | 13 (16) | 20 (25) | 17 (21) | 3 (3) | 4 (4) | 5 (6) | 3 (5)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Energy increased (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 25 (39) | 28 (44) | 28 (50) | 25 (40) | 25 (48) | 26 (35) | 18 (24) | 24 (30) | 18 (28) | 15 (21)
Influenza like illness (General disorders) | 4 (5) | 3 (5) | 4 (7) | 2 (2) | 2 (3) | 3 (4) | 2 (3) | 4 (4) | 1 (1) | 1 (1)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 2 (2) | 4 (4) | 3 (3) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site hypoaesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site lymphadenopathy (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 37 (66) | 42 (75) | 41 (92) | 43 (69) | 42 (76) | 44 (99) | 18 (24) | 22 (28) | 23 (40) | 39 (66)
Injection site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 5 (6) | 4 (4) | 5 (6) | 5 (5) | 4 (4) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site warmth (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 11 (17) | 8 (8) | 9 (10) | 6 (9) | 9 (11) | 5 (6) | 4 (5) | 6 (6) | 6 (7)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (4) | 4 (4) | 2 (3) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 7 (7) | 5 (5) | 4 (6) | 3 (3) | 4 (4) | 5 (6) | 9 (9) | 7 (7) | 4 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte percentage decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte percentage increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil percentage decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 13 (19) | 13 (17) | 6 (6) | 13 (17) | 13 (18) | 7 (8) | 6 (6) | 5 (6) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 24 (37) | 23 (36) | 30 (47) | 27 (33) | 26 (36) | 28 (44) | 10 (12) | 14 (15) | 15 (19) | 12 (17)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periostitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 25 (37) | 29 (50) | 30 (50) | 31 (49) | 25 (42) | 34 (55) | 20 (26) | 25 (43) | 20 (31) | 23 (28)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (3) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 1 (2) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 1 (1) | 5 (7) | 5 (5) | 1 (1) | 5 (5) | 4 (4) | 6 (6) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT03275389/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT03275389/SAP_001.pdf